CLINICAL TRIAL: NCT03928821
Title: A Phase 1 Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of Combinations of Monoclonal Antibodies PGT121, PGDM1400, 10-1074, and VRC07-523LS Administered Via Intravenous Infusion in Healthy, HIV-uninfected Adult Participants
Brief Title: Evaluating the Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of Combinations of Monoclonal Antibodies PGT121, PGDM1400, 10-1074, and VRC07-523LS Administered Via Intravenous Infusion in Healthy, HIV-uninfected Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HVTN 130/HPTN 089; 38531 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2019-04-23; First posted 2019-04-26 (Actual); Results first posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-06

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: PGT121 + VRC07-523LS (Experimental): Participants will receive PGT121 and VRC07-523LS administered sequentially in this order at Day 0.
  Interventions: Biological: PGT121; Biological: VRC07-523LS
- Group 2: PGDM1400 + VRC07-523LS (Experimental): Participants will receive PGDM1400 and VRC07-523LS administered sequentially in this order at Day 0.
  Interventions: Biological: PGDM1400; Biological: VRC07-523LS
- Group 3: 10-1074 + VRC07-523LS (Experimental): Participants will receive 10-1074 and VRC07-523LS administered sequentially in this order at Day 0.
  Interventions: Biological: 10-1074; Biological: VRC07-523LS
- Group 4: PGDM1400 + PGT121 + VRC07-523LS (Experimental): Participants will receive PGDM1400, PGT121, and VRC07-523LS administered sequentially in this order at Day 0 and Month 4.
  Interventions: Biological: PGT121; Biological: PGDM1400; Biological: VRC07-523LS

INTERVENTIONS:
Biological: PGT121 — 20 mg/kg administered intravenously
  Arms: Group 1: PGT121 + VRC07-523LS; Group 4: PGDM1400 + PGT121 + VRC07-523LS
Biological: PGDM1400 — 20 mg/kg administered intravenously
  Arms: Group 2: PGDM1400 + VRC07-523LS; Group 4: PGDM1400 + PGT121 + VRC07-523LS
Biological: 10-1074 — 20 mg/kg administered intravenously
  Arms: Group 3: 10-1074 + VRC07-523LS
Biological: VRC07-523LS — 20 mg/kg administered intravenously

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and antiviral activity of combinations of monoclonal antibodies PGT121, PGDM1400, 10-1074, and VRC07-523LS administered via intravenous infusion in healthy, HIV-uninfected adults.

DETAILED DESCRIPTION:
This study will evaluate the safety, tolerability, pharmacokinetics, and antiviral activity of combinations of monoclonal antibodies PGT121, PGDM1400, 10-1074, and VRC07-523LS administered via intravenous infusion in healthy, HIV-uninfected adults.

Participants will initially be enrolled into one of three groups. At Day 0, Groups 1, 2, and 3 will receive dual combinations of mAbs administered sequentially via IV. Group 1 will receive a combination of PGT121 and VRC07-523LS, Group 2 will receive PGDM1400 and VRC07-523LS, and Group 3 will receive 10-1074 and VRC07-523LS.

Study staff will review study data from Groups 1, 2, and 3 and determine if Group 4 may begin to enroll. Participants in Group 4 will receive PGDM1400, PGT121, and VRC07-523LS administered in sequence via IV on Day 0 and at Month 4.

Study duration will be 12 months for participants in Groups 1, 2, and 3, and 16 months for participants in Group 4. Participants will attend several study visits, which may include physical examinations, blood and urine collection, HIV testing and pretest counseling, risk reduction counseling, and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

General and Demographic Criteria

* Age of 18 to 50 years
* Access to a participating clinical research site (CRS) and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: volunteer demonstrates understanding of this study and completes a questionnaire prior to first study product administration with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Agrees not to enroll in another study of an investigational research agent until completion of the last required protocol clinic visit
* Good general health as shown by medical history, physical exam, and screening laboratory tests

HIV-Related Criteria:

* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks and amenable to HIV risk reduction counseling
* Assessed by the clinic staff as being at "low risk" for HIV infection and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit (see the protocol for more information)

Laboratory Inclusion Values

Hemogram/Complete Blood Count

* Hemoglobin greater than or equal to 11.0 g/dL for volunteers who were assigned female sex at birth, greater than or equal to 13.0 g/dL for volunteers who were assigned male sex at birth. For transgender participants who have been on feminizing hormone therapy for more than 6 consecutive months, determine hemoglobin eligibility based on the gender with which they identify (ie, a transgender female who has been on hormone therapy for more than 6 consecutive months should be assessed for eligibility using the hemoglobin parameters for persons assigned female sex at birth).
* White blood cell count equal to 2,500 to 12,000 cells/mm^3
* White blood cell (WBC) differential either within institutional normal range or with site clinician approval
* Platelets equal to 125,000 to 550,000/mm^3

Chemistry

* Chemistry panel: Alanine aminotransferase (ALT) less than 1.25 times the institutional upper limit of normal; creatinine less than or equal to institutional upper limit of normal

Virology

* Negative HIV-1 and -2 blood test: US volunteers must have a negative Food and Drug Administration (FDA)-approved enzyme immunoassay (EIA) or chemiluminescent microparticle immunoassay (CMIA).
* Negative Hepatitis B surface antigen (HBsAg)
* Negative anti-Hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive

Urine

* Negative or trace urine protein

Reproductive Status

* Volunteers who were assigned female sex at birth: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed prior to study product administration on the day of initial study product administration. Persons who are NOT of reproductive potential due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing.
* Reproductive status: A volunteer who was assigned female sex at birth must:

  * Agree to use effective contraception for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit. Effective contraception is defined as using one of the following methods:
  * Condoms (male or female) with or without a spermicide,
  * Diaphragm or cervical cap with spermicide,
  * Intrauterine device (IUD),
  * Hormonal contraception,
  * Tubal ligation,
  * Any other contraceptive method approved by the HVTN 130/HPTN 089 Protocol Safety Review Team (PSRT)
  * Successful vasectomy in any partner assigned male sex at birth (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity postvasectomy);
  * Or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy or bilateral oophorectomy;
  * Or be sexually abstinent.
* Volunteers who were assigned female sex at birth must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit.

Exclusion Criteria:

General

* Weight greater than 115 kg
* Blood products received within 120 days before first study product administration, unless eligibility for earlier enrollment is determined by the HVTN 130/HPTN 089 PSRT
* Investigational research agents received within 30 days before first study product administration
* Intent to participate in another study of an investigational research agent or any other study that requires non-Network HIV antibody testing during the planned duration of the HVTN 130/HPTN 089 study
* Pregnant or breastfeeding

Vaccines and other Injections

* HIV vaccine(s) received in a prior HIV vaccine trial. For volunteers who have received control/placebo in an HIV vaccine trial, the HVTN 130/HPTN 089 PSRT will determine eligibility on a case-by-case basis.
* Previous receipt of humanized or human mAbs, whether licensed or investigational; the HVTN 130/HPTN 089 PSRT will determine eligibility on a case-by-case basis.
* Previous receipt of monoclonal antibodies VRC01, VRC01LS, VRC07-523LS, PGT121, PGDM1400, or 10-1074

Immune System

* Immunosuppressive medications received within 30 days before first study product administration (Not exclusionary: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatological condition; or [4] a single course of oral/parenteral prednisone or equivalent at doses less than 20 mg/day and length of therapy less than 14 days.)
* Serious adverse reactions to VRC07-523LS, PGT121, PGDM1400, or 10-1074 formulation components (acetate, sucrose, polysorbate 80, histidine, and sorbitol; see the protocol for more information), including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain
* Immunoglobulin received within 90 days before first study product administration, unless eligibility for earlier enrollment is determined by the HVTN 130/HPTN 089 PSRT (for mAb see criterion above)
* Autoimmune disease (Not excluded from participation: Volunteer with mild, stable and uncomplicated autoimmune disease that does not require immunosuppressive medication and that, in the judgment of the site investigator, is likely not subject to exacerbation and likely not to complicate Solicited and Unsolicited AE assessments)
* Immunodeficiency

Clinically significant medical conditions

* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

  * A process that would affect the immune response,
  * A process that would require medication that affects the immune response,
  * Any contraindication to repeated infusions, or blood draws, including inability to establish venous or sub-cutaneous access.
  * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period,
  * A condition or process (eg, chronic urticaria or recent injection or infusion with evidence of residual inflammation) for which signs or symptoms could be confused with reactions to the study product, or
  * Any condition specifically listed among the exclusion criteria.
* Any medical, psychiatric, occupational, or skin condition (eg, tattoos) that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety, Solicited AEs, or a volunteer's ability to give informed consent
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Current anti-tuberculosis (TB) therapy
* Asthma other than mild, well-controlled asthma (Symptoms of asthma severity as defined in the most recent National Asthma Education and Prevention Program (NAEPP) Expert Panel report). Exclude a volunteer who:

  * Uses a short-acting rescue inhaler (typically a beta 2 agonist) daily, or
  * Uses moderate/high-dose, inhaled corticosteroids, or
  * In the past year has had either of the following:
  * Greater than 1 exacerbation of symptoms treated with oral/parenteral corticosteroids;
  * Needed emergency care, urgent care, hospitalization, or intubation for asthma.
* Diabetes mellitus type 1 or type 2 (Not exclusionary: type 2 cases controlled with diet alone or a history of isolated gestational diabetes)
* Hypertension:

  * If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined as consistently less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be less than or equal to 150 mm Hg systolic and less than or equal to 100 mm Hg diastolic. For these volunteers, blood pressure must be less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic at enrollment.
  * If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure greater than or equal to 150 mm Hg at enrollment or diastolic blood pressure greater than or equal to 100 mm Hg at enrollment.
* Bleeding disorder diagnosed by a clinician (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (Not excluded from participation: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study.)
* Seizure disorder: History of seizure(s) within past three years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* Asplenia: any condition resulting in the absence of a functional spleen
* History of hereditary angioedema, acquired angioedema, or idiopathic angioedema

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Sobieszczyk, Study Chair — Columbia University; Sharon Mannheimer, Study Chair — Columbia University
Locations (4):
- United States (4):
  - Fenway Health (FH) CRS, Boston, Massachusetts
  - Harlem Prevention Center CRS, New York, New York
  - Columbia P&S CRS, New York, New York
  - Vanderbilt Vaccine (VV) CRS, Nashville, Tennessee

REFERENCES:
- [Derived] Sobieszczyk ME, Mannheimer S, Paez CA, Yu C, Gamble T, Theodore DA, Chege W, Yacovone M, Hanscom B, Heptinstall J, Seaton KE, Zhang L, Miner MD, Eaton A, Weiner JA, Mayer K, Kalams S, Stephenson K, Julg B, Caskey M, Nussenzweig M, Gama L, Barouch DH, Ackerman ME, Tomaras GD, Huang Y, Montefiori D; HVTN 130/HPTN 089 Study Team. Safety, tolerability, pharmacokinetics, and immunological activity of dual-combinations and triple-combinations of anti-HIV monoclonal antibodies PGT121, PGDM1400, 10-1074, and VRC07-523LS administered intravenously to HIV-uninfected adults: a phase 1 randomised trial. Lancet HIV. 2023 Oct;10(10):e653-e662. doi: 10.1016/S2352-3018(23)00140-6. PMID 37802566

RESULTS

PARTICIPANT FLOW:
Groups:
- T1: PGT121 + VRC07-523LS mo 0: PGT121 20 mg/kg AND VRC07-523LS 20 mg/kg to be administered IV sequentially in this order at Month 0.
- T2: PGDM1400 + VRC07-523LS mo 0: PGDM1400 20 mg/kg AND VRC07-523LS 20 mg/kg to be administered IV sequentially in this order at Month 0.
- T3: 10-1074 + VRC07-523LS: 10-1074 20 mg/kg AND VRC07-523LS 20 mg/kg to be administered IV sequentially in this order at Month 0.
- T4: PGT121 + PGDM1400 + VRC07-523LS mo(0, 4): PGDM1400 20 mg/kg AND PGT121 20 mg/kg AND VRC07-523LS 20 mg/kg to be administered IV sequentially in this order at Month 0 and Month 4.
Period: Overall Study
Arm/Group | T1: PGT121 + VRC07-523LS mo 0 | T2: PGDM1400 + VRC07-523LS mo 0 | T3: 10-1074 + VRC07-523LS | T4: PGT121 + PGDM1400 + VRC07-523LS mo(0, 4)
Started | 6 | 6 | 6 | 9
Completed | 6 | 3 | 3 | 8
Not Completed | 0 | 3 | 3 | 1
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 3 | 0
Not completed — Participant Unable to Adhere to Visit Schedule | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T1: PGT121 + VRC07-523LS mo 0 | T2: PGDM1400 + VRC07-523LS mo 0 | T3: 10-1074 + VRC07-523LS | T4: PGT121 + PGDM1400 + VRC07-523LS mo(0, 4) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 9 | 27
Age, Continuous [Median (Full Range); unit: years] | 25 [21 to 25] | 29 [21 to 50] | 28 [25 to 49] | 30 [19 to 49] | 26 [19 to 50]
Age, Customized [Count of Participants; unit: Participants]
  Less than 18 years | 0 | 0 | 0 | 0 | 0
  18 - 20 years | 0 | 0 | 0 | 1 | 1
  21 - 30 years | 6 | 3 | 4 | 4 | 17
  31 - 40 years | 0 | 2 | 0 | 2 | 4
  41 - 50 years | 0 | 1 | 2 | 2 | 5
  Above 50 years | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 3 | 5 | 16
  Male | 1 | 3 | 3 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 2 | 3
  Not Hispanic or Latino | 6 | 5 | 6 | 7 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 1 | 1 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 0 | 2
  White | 5 | 3 | 4 | 7 | 19
  More than one race | 0 | 1 | 0 | 0 | 1
  Other | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 6 | 9 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms: Pain and/or Tenderness
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [July 2017]. The maximum grade observed for each symptom over the time frame is presented.
Time Frame: Measured through 3 days after each vaccine dose at T1-T3: Day 0 and T4: Days 0, 112
Measure: Count of Participants; unit: Participants
Arm/Group | T1: PGT121 + VRC07-523LS mo 0 | T2: PGDM1400 + VRC07-523LS mo 0 | T3: 10-1074 + VRC07-523LS | T4: PGT121 + PGDM1400 + VRC07-523LS mo(0, 4)
Number analyzed (Participants) | 6 | 6 | 6 | 9
Participants
  None | 5 | 6 | 6 | 7
  Mild | 1 | 0 | 0 | 2
  Moderate | 0 | 0 | 0 | 0
  Severe | 0 | 0 | 0 | 0
  Potentially life-threatening | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms: Erythema and/or Induration
Description: as for outcome 1
Time Frame: Measured through 3 days after each vaccine dose at T1-T3: Day 0 and T4: Days 0, 112
Measure: Count of Participants; unit: Participants
Arm/Group | T1: PGT121 + VRC07-523LS mo 0 | T2: PGDM1400 + VRC07-523LS mo 0 | T3: 10-1074 + VRC07-523LS | T4: PGT121 + PGDM1400 + VRC07-523LS mo(0, 4)
Number analyzed (Participants) | 6 | 6 | 6 | 9
Participants
  Erythema/redness: None | 6 | 6 | 6 | 9
  Erythema/redness: Not Gradable | 0 | 0 | 0 | 0
  Erythema/redness: Gr 1: 2.5 to less than 5 cm dim. | 0 | 0 | 0 | 0
  Erythema/redness: Gr 2: 5 to less than 10 cm dim. | 0 | 0 | 0 | 0
  Erythema/redness: Gr 3: >=10 cm dim. | 0 | 0 | 0 | 0
  Erythema/redness: Gr 3: Complications AE | 0 | 0 | 0 | 0
  Erythema/redness: Gr 4: Complications AE | 0 | 0 | 0 | 0
  Induration/swelling: None | 5 | 6 | 6 | 9
  Induration/swelling: Not Gradable | 1 | 0 | 0 | 0
  Induration/swelling: Gr 1: 2.5 to less than 5 cm dim. | 0 | 0 | 0 | 0
  Induration/swelling: Gr 2: 5 to less than 10 cm dim. | 0 | 0 | 0 | 0
  Induration/swelling: Gr 3: >=10 cm dim. | 0 | 0 | 0 | 0
  Induration/swelling: Gr 3: Complications AE | 0 | 0 | 0 | 0
  Induration/swelling: Gr 4: Complications AE | 0 | 0 | 0 | 0
  Erythema and/or Induration: None | 5 | 6 | 6 | 9
  Erythema and/or Induration: Not Gradable | 1 | 0 | 0 | 0
  Erythema and/or Induration: Gr 1: 2.5 to less than 5 cm dim. | 0 | 0 | 0 | 0
  Erythema and/or Induration: Gr 2: 5 to less than 10 cm dim. | 0 | 0 | 0 | 0
  Erythema and/or Induration: Gr 3: >=10 cm dim. | 0 | 0 | 0 | 0
  Erythema and/or Induration: Gr 3: Complications AE | 0 | 0 | 0 | 0
  Erythema and/or Induration: Gr 4: Complications AE | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [July 2017]. The following symptoms are considered as systemic reactogenicity if the onset date was within the periods of assessment specified in the protocol: malaise and/or fatigue, myalgia, headache, nausea, vomiting, chills, arthralgia, and body temperature. The item Max. Systemic Symptoms is the maximum of the individual systemic reactogenicities excluding body temperature for a participant.
Time Frame: Measured through 3 days after each vaccine dose at T1-T3: Day 0 and T4: Days 0, 112
Measure: Count of Participants; unit: Participants
Arm/Group | T1: PGT121 + VRC07-523LS mo 0 | T2: PGDM1400 + VRC07-523LS mo 0 | T3: 10-1074 + VRC07-523LS | T4: PGT121 + PGDM1400 + VRC07-523LS mo(0, 4)
Number analyzed (Participants) | 6 | 6 | 6 | 9
Participants
  Arthralgia: None | 5 | 5 | 5 | 9
  Arthralgia: Mild | 1 | 1 | 1 | 0
  Arthralgia: Moderate | 0 | 0 | 0 | 0
  Arthralgia: Severe | 0 | 0 | 0 | 0
  Arthralgia: Potentially life-threatening | 0 | 0 | 0 | 0
  Chills: None | 6 | 4 | 6 | 7
  Chills: Mild | 0 | 1 | 0 | 2
  Chills: Moderate | 0 | 1 | 0 | 0
  Chills: Severe | 0 | 0 | 0 | 0
  Chills: Potentially life-threatening | 0 | 0 | 0 | 0
  Facial flushing: None | 6 | 5 | 6 | 9
  Facial flushing: Mild | 0 | 1 | 0 | 0
  Facial flushing: Moderate | 0 | 0 | 0 | 0
  Facial flushing: Severe | 0 | 0 | 0 | 0
  Facial flushing: Potentially life-threatening | 0 | 0 | 0 | 0
  Generalized pruritus: None | 6 | 6 | 5 | 9
  Generalized pruritus: Mild | 0 | 0 | 1 | 0
  Generalized pruritus: Moderate | 0 | 0 | 0 | 0
  Generalized pruritus: Severe | 0 | 0 | 0 | 0
  Generalized pruritus: Potentially life-threatening | 0 | 0 | 0 | 0
  Headache: None | 3 | 4 | 5 | 9
  Headache: Mild | 3 | 2 | 1 | 0
  Headache: Moderate | 0 | 0 | 0 | 0
  Headache: Severe | 0 | 0 | 0 | 0
  Headache: Potentially life-threatening | 0 | 0 | 0 | 0
  Increased body temperature: None | 6 | 6 | 6 | 9
  Increased body temperature: Mild | 0 | 0 | 0 | 0
  Increased body temperature: Moderate | 0 | 0 | 0 | 0
  Increased body temperature: Severe | 0 | 0 | 0 | 0
  Increased body temperature: Potentially life-threatening | 0 | 0 | 0 | 0
  Malaise and/or fatigue: None | 5 | 2 | 4 | 3
  Malaise and/or fatigue: Mild | 1 | 3 | 1 | 5
  Malaise and/or fatigue: Moderate | 0 | 1 | 1 | 1
  Malaise and/or fatigue: Severe | 0 | 0 | 0 | 0
  Malaise and/or fatigue: Potentially life-threatening | 0 | 0 | 0 | 0
  Myalgia: None | 5 | 5 | 6 | 7
  Myalgia: Mild | 0 | 1 | 0 | 2
  Myalgia: Moderate | 1 | 0 | 0 | 0
  Myalgia: Severe | 0 | 0 | 0 | 0
  Myalgia: Potentially life-threatening | 0 | 0 | 0 | 0
  Nausea: None | 6 | 5 | 4 | 9
  Nausea: Mild | 0 | 1 | 2 | 0
  Nausea: Moderate | 0 | 0 | 0 | 0
  Nausea: Severe | 0 | 0 | 0 | 0
  Nausea: Potentially life-threatening | 0 | 0 | 0 | 0
  Non-exertional dyspnea: None | 6 | 6 | 6 | 9
  Non-exertional dyspnea: Mild | 0 | 0 | 0 | 0
  Non-exertional dyspnea: Moderate | 0 | 0 | 0 | 0
  Non-exertional dyspnea: Severe | 0 | 0 | 0 | 0
  Non-exertional dyspnea: Potentially life-threatening | 0 | 0 | 0 | 0
  Non-exertional tachycardia: None | 6 | 6 | 6 | 9
  Non-exertional tachycardia: Mild | 0 | 0 | 0 | 0
  Non-exertional tachycardia: Moderate | 0 | 0 | 0 | 0
  Non-exertional tachycardia: Severe | 0 | 0 | 0 | 0
  Non-exertional tachycardia: Potentially life-threatening | 0 | 0 | 0 | 0
  Unexplained diaphoresis: None | 6 | 6 | 6 | 9
  Unexplained diaphoresis: Mild | 0 | 0 | 0 | 0
  Unexplained diaphoresis: Moderate | 0 | 0 | 0 | 0
  Unexplained diaphoresis: Severe | 0 | 0 | 0 | 0
  Unexplained diaphoresis: Potentially life-threatening | 0 | 0 | 0 | 0
  Urticaria: None | 6 | 6 | 6 | 9
  Urticaria: Mild | 0 | 0 | 0 | 0
  Urticaria: Moderate | 0 | 0 | 0 | 0
  Urticaria: Severe | 0 | 0 | 0 | 0
  Urticaria: Potentially life-threatening | 0 | 0 | 0 | 0
  Max. Systemic Symptoms: None | 3 | 1 | 2 | 3
  Max. Systemic Symptoms: Mild | 2 | 3 | 3 | 5
  Max. Systemic Symptoms: Moderate | 1 | 2 | 1 | 1
  Max. Systemic Symptoms: Severe | 0 | 0 | 0 | 0
  Max. Systemic Symptoms: Potentially life-threatening | 0 | 0 | 0 | 0
  Temperature (C): None | 6 | 6 | 6 | 9
  Temperature (C): Mild | 0 | 0 | 0 | 0
  Temperature (C): Moderate | 0 | 0 | 0 | 0
  Temperature (C): Severe | 0 | 0 | 0 | 0
  Temperature (C): Potentially life-threatening | 0 | 0 | 0 | 0

4. Primary Outcome: Chemistry and Hematology Laboratory Measures - Alanine Aminotransferase (ALT) in U/L
Description: For each local laboratory measure, summary statistics were presented by treatment group and timepoint for the overall population.
Time Frame: Measured during Screening, Days 0, 14, 56, 84*, 112, 140*, 168, 224, 280, 336, 392*, and 448*. Days with * are only available for T4
Population: Overall Number of Participants Analyzed represents participants enrolled and eligible for laboratory assessment. Participants do not have laboratory assessments if they attended the visit but laboratory specimens were not collected, missed the scheduled visit, or terminated participation in the study prior to the scheduled visit.
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | T1: PGT121 + VRC07-523LS mo 0 | T2: PGDM1400 + VRC07-523LS mo 0 | T3: 10-1074 + VRC07-523LS | T4: PGT121 + PGDM1400 + VRC07-523LS mo(0, 4)
Number analyzed (Participants) | 6 | 6 | 6 | 9
U/L
  Alanine Aminotransferase (U/L)-Baseline | 15 [14 to 20] | 14 [12 to 15] | 13 [10 to 17] | 14 [12 to 15]
  Alanine Aminotransferase (U/L)-Day 0 | 14 [8 to 17] | 12 [10 to 17] | 13 [10 to 16] | 14 [10 to 16]
  Alanine Aminotransferase (U/L)-Day 14 | 14 [13 to 15] | 16 [11 to 21] | 11 [10 to 12] | 12 [10 to 16]
  Alanine Aminotransferase (U/L)-Day 56: number analyzed (Participants) | 6 | 6 | 5 | 9
  Alanine Aminotransferase (U/L)-Day 56 | 13 [9 to 19] | 15 [11 to 21] | 20 [12 to 21] | 16 [13 to 17]
  Alanine Aminotransferase (U/L)-Day 84: number analyzed (Participants) | 0 | 0 | 0 | 9
  Alanine Aminotransferase (U/L)-Day 84 |  |  |  | 13 [12 to 15]
  Alanine Aminotransferase (U/L)-Day 112: number analyzed (Participants) | 6 | 5 | 5 | 6
  Alanine Aminotransferase (U/L)-Day 112 | 17 [8 to 23] | 9 [9 to 27] | 16 [14 to 17] | 15 [11 to 15]
  Alanine Aminotransferase (U/L)-Day 140: number analyzed (Participants) | 0 | 0 | 0 | 3
  Alanine Aminotransferase (U/L)-Day 140 |  |  |  | 18 [9 to 20]
  Alanine Aminotransferase (U/L)-Day 168: number analyzed (Participants) | 4 | 3 | 4 | 2
  Alanine Aminotransferase (U/L)-Day 168 | 14 [8 to 24] | 11 [10 to 16] | 17 [16 to 18] | 17 [17 to 17]
  Alanine Aminotransferase (U/L)-Day 224: number analyzed (Participants) | 1 | 1 | 0 | 6
  Alanine Aminotransferase (U/L)-Day 224 | 24 [24 to 24] | 12 [12 to 12] |  | 14 [10 to 15]
  Alanine Aminotransferase (U/L)-Day 280: number analyzed (Participants) | 0 | 1 | 4 | 7
  Alanine Aminotransferase (U/L)-Day 280 |  | 12 [12 to 12] | 13 [11 to 27] | 14 [10 to 17]
  Alanine Aminotransferase (U/L)-Day 336: number analyzed (Participants) | 5 | 2 | 3 | 8
  Alanine Aminotransferase (U/L)-Day 336 | 18 [15 to 22] | 8 [7 to 9] | 14 [13 to 23] | 16 [11 to 19]
  Alanine Aminotransferase (U/L)-Day 392: number analyzed (Participants) | 0 | 0 | 0 | 7
  Alanine Aminotransferase (U/L)-Day 392 |  |  |  | 15 [13 to 18]
  Alanine Aminotransferase (U/L)-Day 448: number analyzed (Participants) | 0 | 0 | 0 | 7
  Alanine Aminotransferase (U/L)-Day 448 |  |  |  | 14 [11 to 18]

5. Primary Outcome: Chemistry and Hematology Laboratory Measures - Creatinine in mg/dL
Description: as for outcome 4
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | T1: PGT121 + VRC07-523LS mo 0 | T2: PGDM1400 + VRC07-523LS mo 0 | T3: 10-1074 + VRC07-523LS | T4: PGT121 + PGDM1400 + VRC07-523LS mo(0, 4)
Number analyzed (Participants) | 6 | 6 | 6 | 9
mg/dL
  Creatinine (mg/dL)-Baseline | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  Creatinine (mg/dL)-Day 0 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  Creatinine (mg/dL)-Day 14 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  Creatinine (mg/dL)-Day 56: number analyzed (Participants) | 6 | 6 | 5 | 9
  Creatinine (mg/dL)-Day 56 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  Creatinine (mg/dL)-Day 84: number analyzed (Participants) | 0 | 0 | 0 | 9
  Creatinine (mg/dL)-Day 84 |  |  |  | 1 [1 to 1]
  Creatinine (mg/dL)-Day 112: number analyzed (Participants) | 6 | 5 | 5 | 6
  Creatinine (mg/dL)-Day 112 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  Creatinine (mg/dL)-Day 140: number analyzed (Participants) | 0 | 0 | 0 | 3
  Creatinine (mg/dL)-Day 140 |  |  |  | 1 [1 to 1]
  Creatinine (mg/dL)-Day 168: number analyzed (Participants) | 4 | 3 | 4 | 2
  Creatinine (mg/dL)-Day 168 | 1 [1 to 1] | 1 [0 to 1] | 1 [1 to 1] | 1 [1 to 1]
  Creatinine (mg/dL)-Day 224: number analyzed (Participants) | 1 | 1 | 0 | 6
  Creatinine (mg/dL)-Day 224 | 1 [1 to 1] | 1 [1 to 1] |  | 1 [1 to 1]
  Creatinine (mg/dL)-Day 280: number analyzed (Participants) | 0 | 1 | 4 | 7
  Creatinine (mg/dL)-Day 280 |  | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  Creatinine (mg/dL)-Day 336: number analyzed (Participants) | 5 | 2 | 3 | 8
  Creatinine (mg/dL)-Day 336 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  Creatinine (mg/dL)-Day 392: number analyzed (Participants) | 0 | 0 | 0 | 7
  Creatinine (mg/dL)-Day 392 |  |  |  | 1 [1 to 1]
  Creatinine (mg/dL)-Day 448: number analyzed (Participants) | 0 | 0 | 0 | 7
  Creatinine (mg/dL)-Day 448 |  |  |  | 1 [1 to 1]

6. Primary Outcome: Chemistry and Hematology Laboratory Measures - Hemoglobin in g/dL
Description: as for outcome 4
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | T1: PGT121 + VRC07-523LS mo 0 | T2: PGDM1400 + VRC07-523LS mo 0 | T3: 10-1074 + VRC07-523LS | T4: PGT121 + PGDM1400 + VRC07-523LS mo(0, 4)
Number analyzed (Participants) | 6 | 6 | 6 | 9
g/dL
  Hemoglobin (g/dL)-Baseline | 14 [13 to 15] | 14 [13 to 14] | 15 [11 to 15] | 14 [13 to 14]
  Hemoglobin (g/dL)-Day 0 | 13 [12 to 15] | 13 [13 to 14] | 13 [11 to 15] | 14 [13 to 14]
  Hemoglobin (g/dL)-Day 14 | 13 [12 to 14] | 14 [13 to 15] | 13 [11 to 14] | 14 [12 to 15]
  Hemoglobin (g/dL)-Day 56: number analyzed (Participants) | 6 | 6 | 5 | 9
  Hemoglobin (g/dL)-Day 56 | 13 [12 to 14] | 14 [13 to 15] | 14 [11 to 14] | 14 [13 to 15]
  Hemoglobin (g/dL)-Day 84: number analyzed (Participants) | 0 | 0 | 0 | 9
  Hemoglobin (g/dL)-Day 84 |  |  |  | 15 [13 to 15]
  Hemoglobin (g/dL)-Day 112: number analyzed (Participants) | 6 | 5 | 5 | 6
  Hemoglobin (g/dL)-Day 112 | 13 [13 to 15] | 13 [13 to 15] | 14 [11 to 14] | 13 [12 to 14]
  Hemoglobin (g/dL)-Day 140: number analyzed (Participants) | 0 | 0 | 0 | 3
  Hemoglobin (g/dL)-Day 140 |  |  |  | 14 [13 to 14]
  Hemoglobin (g/dL)-Day 168: number analyzed (Participants) | 4 | 3 | 4 | 2
  Hemoglobin (g/dL)-Day 168 | 13 [13 to 13] | 13 [13 to 14] | 14 [13 to 15] | 14 [14 to 14]
  Hemoglobin (g/dL)-Day 224: number analyzed (Participants) | 1 | 1 | 0 | 6
  Hemoglobin (g/dL)-Day 224 | 13 [13 to 13] | 13 [13 to 13] |  | 14 [12 to 15]
  Hemoglobin (g/dL)-Day 280: number analyzed (Participants) | 0 | 1 | 4 | 7
  Hemoglobin (g/dL)-Day 280 |  | 13 [13 to 13] | 12 [11 to 14] | 14 [13 to 14]
  Hemoglobin (g/dL)-Day 336: number analyzed (Participants) | 5 | 2 | 3 | 8
  Hemoglobin (g/dL)-Day 336 | 13 [13 to 14] | 13 [12 to 14] | 13 [11 to 14] | 14 [13 to 15]
  Hemoglobin (g/dL)-Day 392: number analyzed (Participants) | 0 | 0 | 0 | 6
  Hemoglobin (g/dL)-Day 392 |  |  |  | 14 [13 to 15]
  Hemoglobin (g/dL)-Day 448: number analyzed (Participants) | 0 | 0 | 0 | 7
  Hemoglobin (g/dL)-Day 448 |  |  |  | 14 [13 to 15]

7. Primary Outcome: Chemistry and Hematology Laboratory Measures - Lymphocyte Count, Neutrophil Count in 1000 Cells/Cubic mm
Description: as for outcome 4
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: 1000 cells/cubic mm
Arm/Group | T1: PGT121 + VRC07-523LS mo 0 | T2: PGDM1400 + VRC07-523LS mo 0 | T3: 10-1074 + VRC07-523LS | T4: PGT121 + PGDM1400 + VRC07-523LS mo(0, 4)
Number analyzed (Participants) | 6 | 6 | 6 | 9
1000 cells/cubic mm
  Lymphocytes (1000 cells/cubic mm)-Baseline | 1.65 [1.33 to 2.13] | 2.191 [1.67 to 2.46] | 1.551 [0.89 to 1.946] | 2.31 [1.48 to 2.605]
  Lymphocytes (1000 cells/cubic mm)-Day 0 | 1.778 [1.13 to 2.18] | 1.785 [1.618 to 2.2] | 1.445 [1.32 to 1.612] | 1.802 [1.68 to 2.17]
  Lymphocytes (1000 cells/cubic mm)-Day 14 | 1.63 [1.3 to 1.719] | 1.781 [1.528 to 1.95] | 1.54 [1.385 to 2.279] | 1.99 [1.58 to 2.69]
  Lymphocytes (1000 cells/cubic mm)-Day 56: number analyzed (Participants) | 6 | 6 | 5 | 9
  Lymphocytes (1000 cells/cubic mm)-Day 56 | 1.824 [1.375 to 1.982] | 1.667 [1.59 to 1.84] | 1.723 [1.36 to 2.033] | 2.176 [1.72 to 2.24]
  Lymphocytes (1000 cells/cubic mm)-Day 84: number analyzed (Participants) | 0 | 0 | 0 | 9
  Lymphocytes (1000 cells/cubic mm)-Day 84 |  |  |  | 1.83 [1.761 to 2.27]
  Lymphocytes (1000 cells/cubic mm)-Day 112: number analyzed (Participants) | 6 | 5 | 5 | 6
  Lymphocytes (1000 cells/cubic mm)-Day 112 | 1.693 [1.2 to 2.255] | 1.768 [1.529 to 1.9] | 1.22 [1.21 to 2.048] | 2.002 [1.55 to 2.14]
  Lymphocytes (1000 cells/cubic mm)-Day 140: number analyzed (Participants) | 0 | 0 | 0 | 3
  Lymphocytes (1000 cells/cubic mm)-Day 140 |  |  |  | 1.487 [1.4 to 1.67]
  Lymphocytes (1000 cells/cubic mm)-Day 168: number analyzed (Participants) | 4 | 3 | 4 | 2
  Lymphocytes (1000 cells/cubic mm)-Day 168 | 1.688 [1.465 to 2.009] | 2.015 [1.97 to 2.42] | 1.918 [1.405 to 2.195] | 1.65 [1.64 to 1.66]
  Lymphocytes (1000 cells/cubic mm)-Day 224: number analyzed (Participants) | 1 | 1 | 0 | 6
  Lymphocytes (1000 cells/cubic mm)-Day 224 | 1.02 [1.02 to 1.02] | 2.9 [2.9 to 2.9] |  | 2.015 [1.5 to 2.16]
  Lymphocytes (1000 cells/cubic mm)-Day 280: number analyzed (Participants) | 0 | 1 | 4 | 7
  Lymphocytes (1000 cells/cubic mm)-Day 280 |  | 2.14 [2.14 to 2.14] | 1.563 [1.32 to 1.93] | 1.74 [1.49 to 2.22]
  Lymphocytes (1000 cells/cubic mm)-Day 336: number analyzed (Participants) | 5 | 2 | 3 | 8
  Lymphocytes (1000 cells/cubic mm)-Day 336 | 1.651 [1.26 to 1.762] | 1.764 [1.72 to 1.807] | 1.927 [1.288 to 2.035] | 1.898 [1.675 to 2.1]
  Lymphocytes (1000 cells/cubic mm)-Day 392: number analyzed (Participants) | 0 | 0 | 0 | 6
  Lymphocytes (1000 cells/cubic mm)-Day 392 |  |  |  | 1.849 [1.74 to 2.15]
  Lymphocytes (1000 cells/cubic mm)-Day 448: number analyzed (Participants) | 0 | 0 | 0 | 7
  Lymphocytes (1000 cells/cubic mm)-Day 448 |  |  |  | 1.76 [1.57 to 2]
  Neutrophils (1000 cells/cubic mm)-Baseline | 3.338 [3.072 to 4.602] | 3.56 [3.227 to 3.71] | 3.39 [2.46 to 3.962] | 4.194 [2.97 to 5.97]
  Neutrophils (1000 cells/cubic mm)-Day 0 | 3.307 [2.616 to 3.91] | 3.032 [2.5 to 3.856] | 2.962 [2.88 to 4.8] | 4.3 [3.42 to 5.32]
  Neutrophils (1000 cells/cubic mm)-Day 14 | 3.181 [2.573 to 3.382] | 4.037 [3.71 to 4.395] | 4.024 [3.135 to 4.73] | 4.831 [3.7 to 5.05]
  Neutrophils (1000 cells/cubic mm)-Day 56: number analyzed (Participants) | 6 | 6 | 5 | 9
  Neutrophils (1000 cells/cubic mm)-Day 56 | 2.762 [2.655 to 3.36] | 3.581 [2.67 to 4.68] | 3.55 [3.235 to 4.082] | 4.98 [4.07 to 5.624]
  Neutrophils (1000 cells/cubic mm)-Day 84: number analyzed (Participants) | 0 | 0 | 0 | 9
  Neutrophils (1000 cells/cubic mm)-Day 84 |  |  |  | 4.12 [3.22 to 5.48]
  Neutrophils (1000 cells/cubic mm)-Day 112: number analyzed (Participants) | 6 | 5 | 5 | 6
  Neutrophils (1000 cells/cubic mm)-Day 112 | 3.377 [2.654 to 3.714] | 3.22 [2.86 to 3.98] | 2.944 [2.39 to 3.66] | 3.735 [2.42 to 4.181]
  Neutrophils (1000 cells/cubic mm)-Day 140: number analyzed (Participants) | 0 | 0 | 0 | 3
  Neutrophils (1000 cells/cubic mm)-Day 140 |  |  |  | 4.108 [2.45 to 4.47]
  Neutrophils (1000 cells/cubic mm)-Day 168: number analyzed (Participants) | 4 | 3 | 4 | 2
  Neutrophils (1000 cells/cubic mm)-Day 168 | 3.882 [3.524 to 4.208] | 4.285 [2.31 to 6.16] | 3.272 [2.662 to 3.479] | 3.155 [2.63 to 3.68]
  Neutrophils (1000 cells/cubic mm)-Day 224: number analyzed (Participants) | 1 | 1 | 0 | 6
  Neutrophils (1000 cells/cubic mm)-Day 224 | 5.24 [5.24 to 5.24] | 3.38 [3.38 to 3.38] |  | 2.855 [2.73 to 4.77]
  Neutrophils (1000 cells/cubic mm)-Day 280: number analyzed (Participants) | 0 | 1 | 4 | 7
  Neutrophils (1000 cells/cubic mm)-Day 280 |  | 3.35 [3.35 to 3.35] | 3.922 [3.112 to 4.357] | 4.14 [2.02 to 5.257]
  Neutrophils (1000 cells/cubic mm)-Day 336: number analyzed (Participants) | 5 | 2 | 3 | 8
  Neutrophils (1000 cells/cubic mm)-Day 336 | 3.93 [2.672 to 3.994] | 2.858 [2.72 to 2.995] | 2.315 [1.9 to 4.752] | 3 [2.88 to 4.868]
  Neutrophils (1000 cells/cubic mm)-Day 392: number analyzed (Participants) | 0 | 0 | 0 | 6
  Neutrophils (1000 cells/cubic mm)-Day 392 |  |  |  | 3.565 [2.68 to 5.25]
  Neutrophils (1000 cells/cubic mm)-Day 448: number analyzed (Participants) | 0 | 0 | 0 | 7
  Neutrophils (1000 cells/cubic mm)-Day 448 |  |  |  | 3.81 [2.99 to 5.491]

8. Primary Outcome: Chemistry and Hematology Laboratory Measures - Platelets, WBC in 1000 Cells/Cubic mm
Description: as for outcome 4
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: 1000 cells/cubic mm
Arm/Group | T1: PGT121 + VRC07-523LS mo 0 | T2: PGDM1400 + VRC07-523LS mo 0 | T3: 10-1074 + VRC07-523LS | T4: PGT121 + PGDM1400 + VRC07-523LS mo(0, 4)
Number analyzed (Participants) | 6 | 6 | 6 | 9
1000 cells/cubic mm
  WBC (1000 cells/cubic mm)-Baseline | 6.25 [5.5 to 7.54] | 6.615 [5.4 to 6.9] | 5.6 [4.63 to 6.4] | 6.1 [5.9 to 9.61]
  WBC (1000 cells/cubic mm)-Day 0 | 6.145 [5.2 to 6.46] | 5.665 [5.33 to 6.8] | 5.4 [4.83 to 6.76] | 6.53 [6.3 to 8.2]
  WBC (1000 cells/cubic mm)-Day 14 | 5.55 [4.9 to 6.34] | 6.645 [5.8 to 6.8] | 6.27 [5.5 to 6.87] | 7.49 [5.9 to 7.7]
  WBC (1000 cells/cubic mm)-Day 56: number analyzed (Participants) | 6 | 6 | 5 | 9
  WBC (1000 cells/cubic mm)-Day 56 | 5.25 [5.1 to 6.5] | 5.985 [5.7 to 7.29] | 5.6 [5.47 to 6.5] | 7.8 [7.6 to 8.6]
  WBC (1000 cells/cubic mm)-Day 84: number analyzed (Participants) | 0 | 0 | 0 | 9
  WBC (1000 cells/cubic mm)-Day 84 |  |  |  | 6.5 [6.3 to 8]
  WBC (1000 cells/cubic mm)-Day 112: number analyzed (Participants) | 6 | 5 | 5 | 6
  WBC (1000 cells/cubic mm)-Day 112 | 5.85 [5.4 to 6.78] | 6.4 [5.2 to 6.76] | 4.9 [4.6 to 6.87] | 6.15 [5.26 to 6.9]
  WBC (1000 cells/cubic mm)-Day 140: number analyzed (Participants) | 0 | 0 | 0 | 3
  WBC (1000 cells/cubic mm)-Day 140 |  |  |  | 6.3 [4.3 to 6.7]
  WBC (1000 cells/cubic mm)-Day 168: number analyzed (Participants) | 4 | 3 | 4 | 2
  WBC (1000 cells/cubic mm)-Day 168 | 6.29 [6.19 to 6.42] | 6.9 [5.77 to 9.15] | 5.35 [5.15 to 5.78] | 5.35 [4.8 to 5.9]
  WBC (1000 cells/cubic mm)-Day 224: number analyzed (Participants) | 1 | 1 | 0 | 6
  WBC (1000 cells/cubic mm)-Day 224 | 6.93 [6.93 to 6.93] | 7.07 [7.07 to 7.07] |  | 5.6 [4.8 to 7.5]
  WBC (1000 cells/cubic mm)-Day 280: number analyzed (Participants) | 0 | 1 | 4 | 7
  WBC (1000 cells/cubic mm)-Day 280 |  | 6.24 [6.24 to 6.24] | 5.9 [5.37 to 6.515] | 6.2 [4.2 to 8.1]
  WBC (1000 cells/cubic mm)-Day 336: number analyzed (Participants) | 5 | 2 | 3 | 8
  WBC (1000 cells/cubic mm)-Day 336 | 5.9 [4.6 to 6.4] | 5.18 [5.06 to 5.3] | 5.1 [3.8 to 7.3] | 5.76 [5.25 to 7.4]
  WBC (1000 cells/cubic mm)-Day 392: number analyzed (Participants) | 0 | 0 | 0 | 6
  WBC (1000 cells/cubic mm)-Day 392 |  |  |  | 6.25 [5.6 to 7]
  WBC (1000 cells/cubic mm)-Day 448: number analyzed (Participants) | 0 | 0 | 0 | 7
  WBC (1000 cells/cubic mm)-Day 448 |  |  |  | 6.2 [5.2 to 7.5]
  Platelets (1000 cells/cubic mm)-Baseline | 219.5 [200 to 259] | 303 [265 to 346] | 245.5 [158 to 299] | 248 [209 to 269]
  Platelets (1000 cells/cubic mm)-Day 0 | 217 [193 to 245] | 317 [244 to 328] | 241.5 [156 to 292] | 267 [246 to 274]
  Platelets (1000 cells/cubic mm)-Day 14 | 218.5 [189 to 242] | 291 [228 to 338] | 244.5 [168 to 314] | 250 [241 to 296]
  Platelets (1000 cells/cubic mm)-Day 56: number analyzed (Participants) | 6 | 6 | 5 | 9
  Platelets (1000 cells/cubic mm)-Day 56 | 228.5 [198 to 242] | 327.5 [258 to 346] | 278 [189 to 346] | 288 [244 to 302]
  Platelets (1000 cells/cubic mm)-Day 84: number analyzed (Participants) | 0 | 0 | 0 | 9
  Platelets (1000 cells/cubic mm)-Day 84 |  |  |  | 259 [250 to 281]
  Platelets (1000 cells/cubic mm)-Day 112: number analyzed (Participants) | 6 | 5 | 5 | 6
  Platelets (1000 cells/cubic mm)-Day 112 | 221.5 [205 to 247] | 349 [272 to 377] | 259 [204 to 297] | 243 [214 to 297]
  Platelets (1000 cells/cubic mm)-Day 140: number analyzed (Participants) | 0 | 0 | 0 | 3
  Platelets (1000 cells/cubic mm)-Day 140 |  |  |  | 195 [174 to 289]
  Platelets (1000 cells/cubic mm)-Day 168: number analyzed (Participants) | 4 | 3 | 4 | 2
  Platelets (1000 cells/cubic mm)-Day 168 | 208 [155.5 to 248] | 380 [265 to 403] | 239 [176 to 301.5] | 159 [127 to 191]
  Platelets (1000 cells/cubic mm)-Day 224: number analyzed (Participants) | 1 | 1 | 0 | 6
  Platelets (1000 cells/cubic mm)-Day 224 | 158 [158 to 158] | 336 [336 to 336] |  | 250.5 [227 to 264]
  Platelets (1000 cells/cubic mm)-Day 280: number analyzed (Participants) | 0 | 1 | 4 | 7
  Platelets (1000 cells/cubic mm)-Day 280 |  | 361 [361 to 361] | 218 [134 to 293] | 254 [234 to 279]
  Platelets (1000 cells/cubic mm)-Day 336: number analyzed (Participants) | 4 | 2 | 3 | 8
  Platelets (1000 cells/cubic mm)-Day 336 | 233 [189 to 258.5] | 373.5 [373 to 374] | 249 [129 to 314] | 242 [234.5 to 267]
  Platelets (1000 cells/cubic mm)-Day 392: number analyzed (Participants) | 0 | 0 | 0 | 6
  Platelets (1000 cells/cubic mm)-Day 392 |  |  |  | 264.5 [212 to 288]
  Platelets (1000 cells/cubic mm)-Day 448: number analyzed (Participants) | 0 | 0 | 0 | 7
  Platelets (1000 cells/cubic mm)-Day 448 |  |  |  | 246 [227 to 296]

9. Primary Outcome: The Number (Percentage) of Participants With Lab Grade > 1 for Alanine Aminotransferase (ALT), Creatinine, Hemoglobin, Lymphocyte Count, Neutrophil Count, Platelets, White Blood Cells (WBC) Was Summarized by Arm
Description: The number (percentage) of participants with lab grade > 1 for alanine aminotransferase (ALT), creatinine, hemoglobin, lymphocyte count, neutrophil count, platelets, white blood cells (WBC) was summarized by arm
Time Frame: Measured during Screening, Days 0, 14, 56, 84*, 112, 140*, 168, 224, 280, 336, 392*, 448*, and 504* Days with * are only available for T4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | T1: PGT121 + VRC07-523LS mo 0 | T2: PGDM1400 + VRC07-523LS mo 0 | T3: 10-1074 + VRC07-523LS | T4: PGT121 + PGDM1400 + VRC07-523LS mo(0, 4)
Number analyzed (Participants) | 6 | 6 | 6 | 9
Participants
  Alanine Aminotransferase (U/L)-Baseline | 0 | 0 | 0 | 0
  Alanine Aminotransferase (U/L)-Day 0 | 0 | 0 | 0 | 0
  Alanine Aminotransferase (U/L)-Day 14 | 0 | 0 | 0 | 0
  Alanine Aminotransferase (U/L)-Day 56: number analyzed (Participants) | 6 | 6 | 5 | 9
  Alanine Aminotransferase (U/L)-Day 56 | 0 | 0 | 0 | 0
  Alanine Aminotransferase (U/L)-Day 84: number analyzed (Participants) | 0 | 0 | 0 | 9
  Alanine Aminotransferase (U/L)-Day 84 | 0 | 0 | 0 | 0
  Alanine Aminotransferase (U/L)-Day 112: number analyzed (Participants) | 6 | 5 | 5 | 6
  Alanine Aminotransferase (U/L)-Day 112 | 0 | 0 | 0 | 0
  Alanine Aminotransferase (U/L)-Day 140: number analyzed (Participants) | 0 | 0 | 0 | 3
  Alanine Aminotransferase (U/L)-Day 140 | 0 | 0 | 0 | 0
  Alanine Aminotransferase (U/L)-Day 168: number analyzed (Participants) | 4 | 3 | 4 | 2
  Alanine Aminotransferase (U/L)-Day 168 | 0 | 0 | 0 | 0
  Alanine Aminotransferase (U/L)-Day 224: number analyzed (Participants) | 1 | 1 | 0 | 6
  Alanine Aminotransferase (U/L)-Day 224 | 0 | 0 | 0 | 0
  Alanine Aminotransferase (U/L)-Day 280: number analyzed (Participants) | 0 | 1 | 4 | 7
  Alanine Aminotransferase (U/L)-Day 280 | 0 | 0 | 0 | 0
  Alanine Aminotransferase (U/L)-Day 336: number analyzed (Participants) | 5 | 2 | 3 | 8
  Alanine Aminotransferase (U/L)-Day 336 | 0 | 0 | 0 | 0
  Alanine Aminotransferase (U/L)-Day 392: number analyzed (Participants) | 0 | 0 | 0 | 7
  Alanine Aminotransferase (U/L)-Day 392 | 0 | 0 | 0 | 0
  Alanine Aminotransferase (U/L)-Day 448: number analyzed (Participants) | 0 | 0 | 0 | 7
  Alanine Aminotransferase (U/L)-Day 448 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)-Baseline | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)-Day 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)-Day 14 | 0 | 0 | 1 | 0
  Hemoglobin (g/dL)-Day 56: number analyzed (Participants) | 6 | 6 | 5 | 9
  Hemoglobin (g/dL)-Day 56 | 0 | 0 | 1 | 0
  Hemoglobin (g/dL)-Day 84: number analyzed (Participants) | 0 | 0 | 0 | 9
  Hemoglobin (g/dL)-Day 84 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)-Day 112: number analyzed (Participants) | 6 | 5 | 5 | 6
  Hemoglobin (g/dL)-Day 112 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)-Day 140: number analyzed (Participants) | 0 | 0 | 0 | 3
  Hemoglobin (g/dL)-Day 140 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)-Day 168: number analyzed (Participants) | 4 | 3 | 4 | 2
  Hemoglobin (g/dL)-Day 168 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)-Day 224: number analyzed (Participants) | 1 | 1 | 0 | 6
  Hemoglobin (g/dL)-Day 224 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)-Day 280: number analyzed (Participants) | 0 | 1 | 4 | 7
  Hemoglobin (g/dL)-Day 280 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)-Day 336: number analyzed (Participants) | 5 | 2 | 3 | 8
  Hemoglobin (g/dL)-Day 336 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)-Day 392: number analyzed (Participants) | 0 | 0 | 0 | 6
  Hemoglobin (g/dL)-Day 392 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)-Day 448: number analyzed (Participants) | 0 | 0 | 0 | 7
  Hemoglobin (g/dL)-Day 448 | 0 | 0 | 0 | 0
  Creatinine (mg/dL)-Baseline | 0 | 0 | 0 | 0
  Creatinine (mg/dL)-Day 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL)-Day 14 | 0 | 0 | 0 | 0
  Creatinine (mg/dL)-Day 56: number analyzed (Participants) | 6 | 6 | 5 | 9
  Creatinine (mg/dL)-Day 56 | 0 | 0 | 0 | 0
  Creatinine (mg/dL)-Day 84: number analyzed (Participants) | 0 | 0 | 0 | 9
  Creatinine (mg/dL)-Day 84 | 0 | 0 | 0 | 0
  Creatinine (mg/dL)-Day 112: number analyzed (Participants) | 6 | 5 | 5 | 6
  Creatinine (mg/dL)-Day 112 | 0 | 0 | 0 | 0
  Creatinine (mg/dL)-Day 140: number analyzed (Participants) | 0 | 0 | 0 | 3
  Creatinine (mg/dL)-Day 140 | 0 | 0 | 0 | 0
  Creatinine (mg/dL)-Day 168: number analyzed (Participants) | 4 | 3 | 4 | 2
  Creatinine (mg/dL)-Day 168 | 0 | 0 | 0 | 0
  Creatinine (mg/dL)-Day 224: number analyzed (Participants) | 1 | 1 | 0 | 6
  Creatinine (mg/dL)-Day 224 | 0 | 0 | 0 | 0
  Creatinine (mg/dL)-Day 280: number analyzed (Participants) | 0 | 1 | 4 | 7
  Creatinine (mg/dL)-Day 280 | 0 | 0 | 0 | 0
  Creatinine (mg/dL)-Day 336: number analyzed (Participants) | 5 | 2 | 3 | 8
  Creatinine (mg/dL)-Day 336 | 0 | 0 | 0 | 0
  Creatinine (mg/dL)-Day 392: number analyzed (Participants) | 0 | 0 | 0 | 7
  Creatinine (mg/dL)-Day 392 | 0 | 0 | 0 | 0
  Creatinine (mg/dL)-Day 448: number analyzed (Participants) | 0 | 0 | 0 | 7
  Creatinine (mg/dL)-Day 448 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm)-Baseline | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm)-Day 0 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm)-Day 14 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm)-Day 56: number analyzed (Participants) | 6 | 6 | 5 | 9
  WBC (1000 cells/cubic mm)-Day 56 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm)-Day 84: number analyzed (Participants) | 0 | 0 | 0 | 9
  WBC (1000 cells/cubic mm)-Day 84 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm)-Day 112: number analyzed (Participants) | 6 | 5 | 5 | 6
  WBC (1000 cells/cubic mm)-Day 112 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm)-Day 140: number analyzed (Participants) | 0 | 0 | 0 | 3
  WBC (1000 cells/cubic mm)-Day 140 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm)-Day 168: number analyzed (Participants) | 4 | 3 | 4 | 2
  WBC (1000 cells/cubic mm)-Day 168 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm)-Day 224: number analyzed (Participants) | 1 | 1 | 0 | 6
  WBC (1000 cells/cubic mm)-Day 224 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm)-Day 280: number analyzed (Participants) | 0 | 1 | 4 | 7
  WBC (1000 cells/cubic mm)-Day 280 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm)-Day 336: number analyzed (Participants) | 5 | 2 | 3 | 8
  WBC (1000 cells/cubic mm)-Day 336 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm)-Day 392: number analyzed (Participants) | 0 | 0 | 0 | 6
  WBC (1000 cells/cubic mm)-Day 392 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm)-Day 448: number analyzed (Participants) | 0 | 0 | 0 | 7
  WBC (1000 cells/cubic mm)-Day 448 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm)-Baseline | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm)-Day 0 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm)-Day 14 | 0 | 0 | 1 | 0
  Platelets (1000 cells/cubic mm)-Day 56: number analyzed (Participants) | 6 | 6 | 5 | 9
  Platelets (1000 cells/cubic mm)-Day 56 | 1 | 0 | 0 | 1
  Platelets (1000 cells/cubic mm)-Day 84: number analyzed (Participants) | 0 | 0 | 0 | 9
  Platelets (1000 cells/cubic mm)-Day 84 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm)-Day 112: number analyzed (Participants) | 6 | 5 | 5 | 6
  Platelets (1000 cells/cubic mm)-Day 112 | 2 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm)-Day 140: number analyzed (Participants) | 0 | 0 | 0 | 3
  Platelets (1000 cells/cubic mm)-Day 140 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm)-Day 168: number analyzed (Participants) | 4 | 3 | 4 | 2
  Platelets (1000 cells/cubic mm)-Day 168 | 1 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm)-Day 224: number analyzed (Participants) | 1 | 1 | 0 | 6
  Platelets (1000 cells/cubic mm)-Day 224 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm)-Day 280: number analyzed (Participants) | 0 | 1 | 4 | 7
  Platelets (1000 cells/cubic mm)-Day 280 | 0 | 0 | 1 | 0
  Platelets (1000 cells/cubic mm)-Day 336: number analyzed (Participants) | 4 | 2 | 3 | 8
  Platelets (1000 cells/cubic mm)-Day 336 | 0 | 0 | 0 | 1
  Platelets (1000 cells/cubic mm)-Day 392: number analyzed (Participants) | 0 | 0 | 0 | 6
  Platelets (1000 cells/cubic mm)-Day 392 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm)-Day 448: number analyzed (Participants) | 0 | 0 | 0 | 7
  Platelets (1000 cells/cubic mm)-Day 448 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm)-Baseline | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm)-Day 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm)-Day 14 | 0 | 0 | 0 | 2
  Lymphocytes (1000 cells/cubic mm)-Day 56: number analyzed (Participants) | 6 | 6 | 5 | 9
  Lymphocytes (1000 cells/cubic mm)-Day 56 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm)-Day 84: number analyzed (Participants) | 0 | 0 | 0 | 9
  Lymphocytes (1000 cells/cubic mm)-Day 84 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm)-Day 112: number analyzed (Participants) | 6 | 5 | 5 | 6
  Lymphocytes (1000 cells/cubic mm)-Day 112 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm)-Day 140: number analyzed (Participants) | 0 | 0 | 0 | 3
  Lymphocytes (1000 cells/cubic mm)-Day 140 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm)-Day 168: number analyzed (Participants) | 4 | 3 | 4 | 2
  Lymphocytes (1000 cells/cubic mm)-Day 168 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm)-Day 224: number analyzed (Participants) | 1 | 1 | 0 | 6
  Lymphocytes (1000 cells/cubic mm)-Day 224 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm)-Day 280: number analyzed (Participants) | 0 | 1 | 4 | 7
  Lymphocytes (1000 cells/cubic mm)-Day 280 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm)-Day 336: number analyzed (Participants) | 5 | 2 | 3 | 8
  Lymphocytes (1000 cells/cubic mm)-Day 336 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm)-Day 392: number analyzed (Participants) | 0 | 0 | 0 | 6
  Lymphocytes (1000 cells/cubic mm)-Day 392 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm)-Day 448: number analyzed (Participants) | 0 | 0 | 0 | 7
  Lymphocytes (1000 cells/cubic mm)-Day 448 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm)-Baseline | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm)-Day 0 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm)-Day 14 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm)-Day 56: number analyzed (Participants) | 6 | 6 | 5 | 9
  Neutrophils (1000 cells/cubic mm)-Day 56 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm)-Day 84: number analyzed (Participants) | 0 | 0 | 0 | 9
  Neutrophils (1000 cells/cubic mm)-Day 84 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm)-Day 112: number analyzed (Participants) | 6 | 5 | 5 | 6
  Neutrophils (1000 cells/cubic mm)-Day 112 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm)-Day 140: number analyzed (Participants) | 0 | 0 | 0 | 3
  Neutrophils (1000 cells/cubic mm)-Day 140 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm)-Day 168: number analyzed (Participants) | 4 | 3 | 4 | 2
  Neutrophils (1000 cells/cubic mm)-Day 168 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm)-Day 224: number analyzed (Participants) | 1 | 1 | 0 | 6
  Neutrophils (1000 cells/cubic mm)-Day 224 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm)-Day 280: number analyzed (Participants) | 0 | 1 | 4 | 7
  Neutrophils (1000 cells/cubic mm)-Day 280 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm)-Day 336: number analyzed (Participants) | 5 | 2 | 3 | 8
  Neutrophils (1000 cells/cubic mm)-Day 336 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm)-Day 392: number analyzed (Participants) | 0 | 0 | 0 | 6
  Neutrophils (1000 cells/cubic mm)-Day 392 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm)-Day 448: number analyzed (Participants) | 0 | 0 | 0 | 7
  Neutrophils (1000 cells/cubic mm)-Day 448 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Participants With Early Discontinuation of Vaccinations and Reason for Discontinuation
Description: The number (percentage) of participants with early discontinuation of vaccinations and reason for discontinuation was summarized by arm. The three participants discontinued treatment in T4 were due to the COVID-19 pandemic lockdown.
Time Frame: Measured through Month 4
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | T1: PGT121 + VRC07-523LS mo 0 | T2: PGDM1400 + VRC07-523LS mo 0 | T3: 10-1074 + VRC07-523LS | T4: PGT121 + PGDM1400 + VRC07-523LS mo(0, 4)
Number analyzed (Participants) | 6 | 6 | 6 | 9
Participants
  Pregnancy | 0 | 0 | 0 | 0
  HIV infection | 0 | 0 | 0 | 0
  Death | 0 | 0 | 0 | 0
  Clinical event other than reactogenicity, HIV infection, or death | 0 | 0 | 0 | 0
  Solicited adverse event symptom | 0 | 0 | 0 | 0
  Investigator Reason | 0 | 0 | 0 | 0
  Participant refused SPA | 0 | 0 | 0 | 0
  Co-Enrollment in a study with an investigational research agent | 0 | 0 | 0 | 0
  Psychiatric reason | 0 | 0 | 0 | 0
  Participant unable to schedule visit within window | 0 | 0 | 0 | 0
  Unable to contact participant | 0 | 0 | 0 | 0
  Incarceration | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 3
  Did not Discontinue SPA | 6 | 6 | 6 | 6

11. Secondary Outcome: Serum Concentration Levels of PGT121, PGDM1400, and VRC07-523LS Among Participants Who Received All Scheduled Product Administrations
Description: Serum PGDM1400, PGT121, and VRC07-523LS IgG levels were measured on a Bio-Plex instrument (Bio-Rad) using a validated assay designed to simultaneously measure infused PGDM1400, PGT121, and VRC07-523LS by its ability to bind anti-idiotype antibody captured on fluorescent magnetic beads. This assay was derived from a standardized custom HIV-1 Luminex assay. PGDM1400, PGT121 and VRC07-523LS were titrated and combined to create a standard curve that was used to determine concentration of the diluted samples. The negative controls were CH58 (an irrelevant mAb) and blank beads.Serum 10-1074 level was measured by anti-idotypic ELISA. Participant serum sample was incubated in anti-ID coated micro-plate well. A conjugated secondary antibody was used to detect bound 10-1074. Samples were titrated to ensure positive optical density (O.D.) readouts fall within the linear range of the assay for monoclonal antibody concentration calculations.
Time Frame: Measured during Screening, Days 0, 3, 6, 14, 28, 56, 84*, 112, 140*, 168, 224, 280, 336, 392*, and 448* Days with * are only available for T4
Population: T1-T3 particiants who received infusion at Day 0 and T4 participants who received infusions at Day 0 and 112 with available serum concentration data. Visits with 0 participants analyzed are due to: (1) mAbs were only assayed for the treatment arms that received those mAbs. (2) Treatment group T4 had more scheduled sample collection visits than treatment groups T1-T3. (3) Data were excluded if the participant didn't receive all scheduled administrations.
Measure: Median (Inter-Quartile Range); unit: mg/ml
Arm/Group | T1: PGT121 + VRC07-523LS mo 0 | T2: PGDM1400 + VRC07-523LS mo 0 | T3: 10-1074 + VRC07-523LS | T4: PGT121 + PGDM1400 + VRC07-523LS mo(0, 4)
Number analyzed (Participants) | 6 | 6 | 6 | 9
mg/ml
  10-1074 (Day- 0): number analyzed (Participants) | 0 | 0 | 5 | 0
  10-1074 (Day- 0) |  |  | 0.21 [0.21 to 0.21] |
  10-1074 (Day- 3): number analyzed (Participants) | 0 | 0 | 5 | 0
  10-1074 (Day- 3) |  |  | 598.55 [444.43 to 844.87] |
  10-1074 (Day- 6): number analyzed (Participants) | 0 | 0 | 5 | 0
  10-1074 (Day- 6) |  |  | 453.99 [378.63 to 529.19] |
  10-1074 (Day- 14): number analyzed (Participants) | 0 | 0 | 5 | 0
  10-1074 (Day- 14) |  |  | 300.15 [279.57 to 315.65] |
  10-1074 (Day- 28): number analyzed (Participants) | 0 | 0 | 5 | 0
  10-1074 (Day- 28) |  |  | 242.22 [140.97 to 253.34] |
  10-1074 (Day- 56): number analyzed (Participants) | 0 | 0 | 4 | 0
  10-1074 (Day- 56) |  |  | 111.62 [81.11 to 127.39] |
  10-1074 (Day-112): number analyzed (Participants) | 0 | 0 | 4 | 0
  10-1074 (Day-112) |  |  | 25.18 [19.22 to 32.51] |
  10-1074 (Day-168): number analyzed (Participants) | 0 | 0 | 4 | 0
  10-1074 (Day-168) |  |  | 8.60 [6.27 to 11.17] |
  10-1074 (Day-224): number analyzed (Participants) | 0 | 0 | 0 | 0
  10-1074 (Day-280): number analyzed (Participants) | 0 | 0 | 3 | 0
  10-1074 (Day-280) |  |  | 0.98 [0.59 to 3.25] |
  10-1074 (Day-336): number analyzed (Participants) | 0 | 0 | 2 | 0
  10-1074 (Day-336) |  |  | 2.44 [1.32 to 3.55] |
  PGDM1400 (Day- 0): number analyzed (Participants) | 0 | 6 | 0 | 6
  PGDM1400 (Day- 0) |  | 0.02 [0.02 to 0.02] |  | 0.02 [0.02 to 0.02]
  PGDM1400 (Day- 3): number analyzed (Participants) | 0 | 6 | 0 | 6
  PGDM1400 (Day- 3) |  | 251.54 [234.47 to 273.48] |  | 209.25 [191.70 to 315.97]
  PGDM1400 (Day- 6): number analyzed (Participants) | 0 | 6 | 0 | 6
  PGDM1400 (Day- 6) |  | 182.23 [160.51 to 186.36] |  | 172.18 [163.04 to 193.95]
  PGDM1400 (Day- 14): number analyzed (Participants) | 0 | 6 | 0 | 6
  PGDM1400 (Day- 14) |  | 139.77 [134.94 to 146.76] |  | 129.97 [116.59 to 143.36]
  PGDM1400 (Day- 28): number analyzed (Participants) | 0 | 6 | 0 | 6
  PGDM1400 (Day- 28) |  | 70.92 [67.17 to 73.87] |  | 67.59 [55.45 to 75.91]
  PGDM1400 (Day- 56): number analyzed (Participants) | 0 | 6 | 0 | 6
  PGDM1400 (Day- 56) |  | 27.88 [26.68 to 31.56] |  | 28.38 [18.02 to 39.50]
  PGDM1400 (Day- 84): number analyzed (Participants) | 0 | 0 | 0 | 6
  PGDM1400 (Day- 84) |  |  |  | 10.93 [7.79 to 14.97]
  PGDM1400 (Day-112): number analyzed (Participants) | 0 | 5 | 0 | 6
  PGDM1400 (Day-112) |  | 5.50 [4.63 to 6.04] |  | 4.99 [3.81 to 7.11]
  PGDM1400 (Day-140): number analyzed (Participants) | 0 | 0 | 0 | 1
  PGDM1400 (Day-140) |  |  |  | 46.07 [46.07 to 46.07]
  PGDM1400 (Day-168): number analyzed (Participants) | 0 | 4 | 0 | 0
  PGDM1400 (Day-168) |  | 1.08 [1.02 to 1.10] |  |
  PGDM1400 (Day-224): number analyzed (Participants) | 0 | 1 | 0 | 3
  PGDM1400 (Day-224) |  | 0.26 [0.26 to 0.26] |  | 6.24 [4.22 to 9.12]
  PGDM1400 (Day-280): number analyzed (Participants) | 0 | 1 | 0 | 5
  PGDM1400 (Day-280) |  | 0.09 [0.09 to 0.09] |  | 1.27 [0.50 to 1.55]
  PGDM1400 (Day-336): number analyzed (Participants) | 0 | 2 | 0 | 6
  PGDM1400 (Day-336) |  | 0.02 [0.02 to 0.02] |  | 0.52 [0.18 to 0.67]
  PGDM1400 (Day-392): number analyzed (Participants) | 0 | 0 | 0 | 5
  PGDM1400 (Day-392) |  |  |  | 0.11 [0.04 to 0.12]
  PGDM1400 (Day-448): number analyzed (Participants) | 0 | 0 | 0 | 5
  PGDM1400 (Day-448) |  |  |  | 0.02 [0.02 to 0.04]
  PGT121 (Day- 0): number analyzed (Participants) | 6 | 0 | 0 | 6
  PGT121 (Day- 0) | 0.05 [0.05 to 0.05] |  |  | 0.05 [0.05 to 0.05]
  PGT121 (Day- 3): number analyzed (Participants) | 6 | 0 | 0 | 6
  PGT121 (Day- 3) | 196.57 [172.85 to 210.31] |  |  | 169.62 [153.15 to 218.39]
  PGT121 (Day- 6): number analyzed (Participants) | 6 | 0 | 0 | 6
  PGT121 (Day- 6) | 129.35 [116.95 to 137.34] |  |  | 130.33 [128.40 to 139.89]
  PGT121 (Day- 14): number analyzed (Participants) | 6 | 0 | 0 | 6
  PGT121 (Day- 14) | 80.12 [79.07 to 86.22] |  |  | 95.54 [90.48 to 101.27]
  PGT121 (Day- 28): number analyzed (Participants) | 6 | 0 | 0 | 6
  PGT121 (Day- 28) | 44.46 [40.81 to 50.03] |  |  | 60.62 [54.15 to 68.21]
  PGT121 (Day- 56): number analyzed (Participants) | 6 | 0 | 0 | 6
  PGT121 (Day- 56) | 22.08 [18.83 to 23.24] |  |  | 25.79 [16.64 to 30.72]
  PGT121 (Day- 84): number analyzed (Participants) | 0 | 0 | 0 | 6
  PGT121 (Day- 84) |  |  |  | 12.42 [9.09 to 15.18]
  PGT121 (Day-112): number analyzed (Participants) | 6 | 0 | 0 | 6
  PGT121 (Day-112) | 4.03 [3.45 to 5.97] |  |  | 5.82 [5.60 to 10.02]
  PGT121 (Day-140): number analyzed (Participants) | 0 | 0 | 0 | 1
  PGT121 (Day-140) |  |  |  | 49.17 [49.17 to 49.17]
  PGT121 (Day-168): number analyzed (Participants) | 4 | 0 | 0 | 0
  PGT121 (Day-168) | 1.70 [0.88 to 3.28] |  |  |
  PGT121 (Day-224): number analyzed (Participants) | 1 | 0 | 0 | 3
  PGT121 (Day-224) | 0.31 [0.31 to 0.31] |  |  | 11.28 [7.72 to 12.63]
  PGT121 (Day-280): number analyzed (Participants) | 0 | 0 | 0 | 5
  PGT121 (Day-280) |  |  |  | 2.36 [1.46 to 4.57]
  PGT121 (Day-336): number analyzed (Participants) | 5 | 0 | 0 | 6
  PGT121 (Day-336) | 0.05 [0.05 to 0.11] |  |  | 1.05 [0.56 to 2.06]
  PGT121 (Day-392): number analyzed (Participants) | 0 | 0 | 0 | 5
  PGT121 (Day-392) |  |  |  | 0.33 [0.17 to 0.65]
  PGT121 (Day-448): number analyzed (Participants) | 0 | 0 | 0 | 5
  PGT121 (Day-448) |  |  |  | 0.10 [0.05 to 0.29]
  VRC07-523LS (Day- 0): number analyzed (Participants) | 6 | 6 | 5 | 6
  VRC07-523LS (Day- 0) | 0.01 [0.01 to 0.02] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.01]
  VRC07-523LS (Day- 3): number analyzed (Participants) | 6 | 6 | 5 | 6
  VRC07-523LS (Day- 3) | 265.97 [262.58 to 300.62] | 239.32 [224.13 to 264.34] | 182.66 [164.80 to 187.40] | 212.11 [195.83 to 306.56]
  VRC07-523LS (Day- 6): number analyzed (Participants) | 6 | 6 | 5 | 6
  VRC07-523LS (Day- 6) | 171.02 [158.01 to 209.24] | 176.51 [158.50 to 183.85] | 176.01 [167.23 to 176.82] | 156.15 [154.76 to 175.84]
  VRC07-523LS (Day- 14): number analyzed (Participants) | 6 | 6 | 5 | 6
  VRC07-523LS (Day- 14) | 134.44 [128.24 to 135.66] | 139.18 [105.71 to 155.86] | 119.67 [90.44 to 145.10] | 140.86 [123.89 to 162.85]
  VRC07-523LS (Day- 28): number analyzed (Participants) | 6 | 6 | 5 | 6
  VRC07-523LS (Day- 28) | 94.58 [88.61 to 102.26] | 96.17 [83.80 to 110.65] | 87.91 [85.13 to 96.66] | 101.42 [97.05 to 107.31]
  VRC07-523LS (Day- 56): number analyzed (Participants) | 6 | 6 | 4 | 6
  VRC07-523LS (Day- 56) | 60.53 [55.78 to 62.70] | 56.91 [56.03 to 58.35] | 59.33 [51.36 to 63.18] | 56.94 [42.61 to 63.36]
  VRC07-523LS (Day- 84): number analyzed (Participants) | 0 | 0 | 0 | 6
  VRC07-523LS (Day- 84) |  |  |  | 39.57 [28.79 to 45.09]
  VRC07-523LS (Day-112): number analyzed (Participants) | 6 | 5 | 4 | 6
  VRC07-523LS (Day-112) | 24.93 [20.69 to 26.88] | 31.65 [20.09 to 33.07] | 29.37 [24.02 to 30.69] | 26.07 [19.85 to 33.70]
  VRC07-523LS (Day-140): number analyzed (Participants) | 0 | 0 | 0 | 1
  VRC07-523LS (Day-140) |  |  |  | 76.03 [76.03 to 76.03]
  VRC07-523LS (Day-168): number analyzed (Participants) | 4 | 4 | 4 | 0
  VRC07-523LS (Day-168) | 14.45 [12.37 to 16.66] | 12.57 [10.74 to 14.17] | 11.57 [9.73 to 12.35] |
  VRC07-523LS (Day-224): number analyzed (Participants) | 1 | 1 | 0 | 3
  VRC07-523LS (Day-224) | 8.47 [8.47 to 8.47] | 11.24 [11.24 to 11.24] |  | 39.86 [31.26 to 42.29]
  VRC07-523LS (Day-280): number analyzed (Participants) | 0 | 1 | 3 | 5
  VRC07-523LS (Day-280) |  | 3.88 [3.88 to 3.88] | 3.17 [1.81 to 3.50] | 15.13 [14.85 to 16.50]
  VRC07-523LS (Day-336): number analyzed (Participants) | 5 | 2 | 3 | 6
  VRC07-523LS (Day-336) | 1.33 [1.08 to 1.38] | 1.31 [1.16 to 1.46] | 1.48 [0.85 to 2.34] | 9.52 [6.85 to 10.98]
  VRC07-523LS (Day-392): number analyzed (Participants) | 0 | 0 | 0 | 5
  VRC07-523LS (Day-392) |  |  |  | 4.49 [2.73 to 5.51]
  VRC07-523LS (Day-448): number analyzed (Participants) | 0 | 0 | 0 | 5
  VRC07-523LS (Day-448) |  |  |  | 2.16 [1.10 to 2.59]

12. Secondary Outcome: Magnitudes of TZM-bl Cells Responses Against mAb-specific Env-pseudotyped Viruses Among Participants Who Received All Scheduled Product Administrations
Description: Neutralizing antibodies against HIV-1 were measured as a function of reductions in Tat-regulated luciferase (Luc) reporter gene expression in TZM-bl cells. The assay performed in TZM-bl cells measured neutralization titers against the Env-pseudotyped viruses sensitive to the bnAbs (i.e., bnAb-specific viruses) in each infusion group.
Time Frame: Measured during Screening, Days 0, 3, 28, 56, 112, 140*, 168*, 224* Days with * are only available for T4
Population: T1-T3 particiants who received infusion at Day 0 and T4 participants who received infusions at Day 0 and 112 with available neutralizing antibody data. Visits with 0 participants are due to: (1) Isolates were mAb-specific and only assayed for the treatment arms that received the specific mAbs. (2) Treatment group T4 had more scheduled sample collection visits than treatment groups T1-T3. (3) Data were excluded if the participant didn't receive all scheduled administrations.
Measure: Median (Inter-Quartile Range); unit: Relative luminescence units (RLU)
Arm/Group | T1: PGT121 + VRC07-523LS mo 0 | T2: PGDM1400 + VRC07-523LS mo 0 | T3: 10-1074 + VRC07-523LS | T4: PGT121 + PGDM1400 + VRC07-523LS mo(0, 4)
Number analyzed (Participants) | 6 | 6 | 6 | 9
Relative luminescence units (RLU)
  6540.v4.c1 (Day- 0): number analyzed (Participants) | 0 | 0 | 0 | 6
  6540.v4.c1 (Day- 0) |  |  |  | 5.00 [5.00 to 5.00]
  6540.v4.c1 (Day- 3): number analyzed (Participants) | 0 | 0 | 0 | 6
  6540.v4.c1 (Day- 3) |  |  |  | 12301.30 [9796.41 to 17398.1]
  6540.v4.c1 (Day- 28): number analyzed (Participants) | 0 | 0 | 0 | 6
  6540.v4.c1 (Day- 28) |  |  |  | 2365.28 [1930.73 to 2730.45]
  6540.v4.c1 (Day- 56): number analyzed (Participants) | 0 | 0 | 0 | 6
  6540.v4.c1 (Day- 56) |  |  |  | 674.62 [512.44 to 784.11]
  6540.v4.c1 (Day-112): number analyzed (Participants) | 0 | 0 | 0 | 6
  6540.v4.c1 (Day-112) |  |  |  | 82.11 [61.03 to 98.13]
  6540.v4.c1 (Day-140): number analyzed (Participants) | 0 | 0 | 0 | 1
  6540.v4.c1 (Day-140) |  |  |  | 1255.62 [1255.62 to 1255.62]
  6540.v4.c1 (Day-168): number analyzed (Participants) | 0 | 0 | 0 | 0
  6540.v4.c1 (Day-224): number analyzed (Participants) | 0 | 0 | 0 | 3
  6540.v4.c1 (Day-224) |  |  |  | 64.76 [46.21 to 113.02]
  CH505TF.N334S.N160A.N280D.1 (Day- 0): number analyzed (Participants) | 0 | 0 | 0 | 6
  CH505TF.N334S.N160A.N280D.1 (Day- 0) |  |  |  | 5.00 [5.00 to 5.00]
  CH505TF.N334S.N160A.N280D.1 (Day- 3): number analyzed (Participants) | 0 | 0 | 0 | 6
  CH505TF.N334S.N160A.N280D.1 (Day- 3) |  |  |  | 13209.26 [9855.80 to 16397.4]
  CH505TF.N334S.N160A.N280D.1 (Day- 28): number analyzed (Participants) | 0 | 0 | 0 | 6
  CH505TF.N334S.N160A.N280D.1 (Day- 28) |  |  |  | 3344.91 [2579.95 to 3806.03]
  CH505TF.N334S.N160A.N280D.1 (Day- 56): number analyzed (Participants) | 0 | 0 | 0 | 6
  CH505TF.N334S.N160A.N280D.1 (Day- 56) |  |  |  | 1491.45 [901.81 to 1966.97]
  CH505TF.N334S.N160A.N280D.1 (Day-112): number analyzed (Participants) | 0 | 0 | 0 | 6
  CH505TF.N334S.N160A.N280D.1 (Day-112) |  |  |  | 339.83 [296.59 to 554.03]
  CH505TF.N334S.N160A.N280D.1 (Day-140): number analyzed (Participants) | 0 | 0 | 0 | 1
  CH505TF.N334S.N160A.N280D.1 (Day-140) |  |  |  | 2563.08 [2563.08 to 2563.08]
  CH505TF.N334S.N160A.N280D.1 (Day-168): number analyzed (Participants) | 0 | 0 | 0 | 0
  CH505TF.N334S.N160A.N280D.1 (Day-224): number analyzed (Participants) | 0 | 0 | 0 | 3
  CH505TF.N334S.N160A.N280D.1 (Day-224) |  |  |  | 429.44 [318.03 to 585.79]
  CNE55.N160K (Day- 0): number analyzed (Participants) | 6 | 6 | 5 | 6
  CNE55.N160K (Day- 0) | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  CNE55.N160K (Day- 3): number analyzed (Participants) | 6 | 6 | 5 | 6
  CNE55.N160K (Day- 3) | 917.25 [686.59 to 1286.70] | 816.88 [725.91 to 847.67] | 493.12 [383.85 to 549.58] | 469.12 [432.41 to 868.21]
  CNE55.N160K (Day- 28): number analyzed (Participants) | 6 | 6 | 5 | 6
  CNE55.N160K (Day- 28) | 259.58 [212.45 to 323.50] | 188.55 [161.50 to 208.80] | 206.12 [171.05 to 268.36] | 218.32 [169.74 to 257.46]
  CNE55.N160K (Day- 56): number analyzed (Participants) | 6 | 6 | 4 | 6
  CNE55.N160K (Day- 56) | 105.02 [91.83 to 118.53] | 91.57 [80.40 to 117.12] | 170.55 [138.00 to 193.64] | 131.99 [106.91 to 149.44]
  CNE55.N160K (Day-112): number analyzed (Participants) | 6 | 5 | 4 | 6
  CNE55.N160K (Day-112) | 28.65 [25.10 to 36.11] | 10.00 [10.00 to 20.95] | 53.48 [38.18 to 59.63] | 47.57 [30.49 to 65.17]
  CNE55.N160K (Day-140): number analyzed (Participants) | 0 | 0 | 0 | 1
  CNE55.N160K (Day-140) |  |  |  | 92.76 [92.76 to 92.76]
  CNE55.N160K (Day-168): number analyzed (Participants) | 0 | 0 | 0 | 0
  CNE55.N160K (Day-224): number analyzed (Participants) | 0 | 0 | 0 | 3
  CNE55.N160K (Day-224) |  |  |  | 58.52 [48.16 to 82.07]
  T250-4 (Day- 0): number analyzed (Participants) | 6 | 6 | 5 | 0
  T250-4 (Day- 0) | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] |
  T250-4 (Day- 3): number analyzed (Participants) | 6 | 6 | 5 | 0
  T250-4 (Day- 3) | 32029.39 [28181.95 to 41032.5] | 91301.02 [79640.01 to 114904.] | 39113.31 [31644.98 to 45736.7] |
  T250-4 (Day- 28): number analyzed (Participants) | 6 | 6 | 5 | 0
  T250-4 (Day- 28) | 6458.16 [5518.54 to 7452.56] | 27318.99 [23401.71 to 30312.3] | 13028.85 [11586.88 to 14345.8] |
  T250-4 (Day- 56): number analyzed (Participants) | 6 | 6 | 4 | 0
  T250-4 (Day- 56) | 2016.84 [1800.34 to 2646.68] | 7523.58 [6020.17 to 8716.04] | 7070.48 [5359.84 to 7736.68] |
  T250-4 (Day-112): number analyzed (Participants) | 6 | 5 | 4 | 0
  T250-4 (Day-112) | 300.37 [266.45 to 650.96] | 800.00 [618.17 to 837.77] | 1189.03 [760.30 to 1712.31] |

13. Secondary Outcome: Serum Concentrations of PGT121, PGDM1400, 10-1074, and VRC07-523LS for All Participants
Description: as for outcome 11
Time Frame: as for outcome 11
Population: All participants enrolled with available serum concentration data. Visits with 0 participants are due to: (1) mAbs were only assayed for the treatment arms that received those mAbs. (2) Treatment group T4 had more scheduled sample collection visits than treatment groups T1-T3.
Measure: Median (Inter-Quartile Range); unit: mg/ml
Arm/Group | T1: PGT121 + VRC07-523LS mo 0 | T2: PGDM1400 + VRC07-523LS mo 0 | T3: 10-1074 + VRC07-523LS | T4: PGT121 + PGDM1400 + VRC07-523LS mo(0, 4)
Number analyzed (Participants) | 6 | 6 | 6 | 9
mg/ml
  10-1074 (Day- 0): number analyzed (Participants) | 0 | 0 | 6 | 0
  10-1074 (Day- 0) |  |  | 0.21 [0.21 to 0.21] |
  10-1074 (Day- 3): number analyzed (Participants) | 0 | 0 | 6 | 0
  10-1074 (Day- 3) |  |  | 521.49 [422.63 to 783.29] |
  10-1074 (Day- 6): number analyzed (Participants) | 0 | 0 | 6 | 0
  10-1074 (Day- 6) |  |  | 416.31 [298.03 to 510.39] |
  10-1074 (Day- 14): number analyzed (Participants) | 0 | 0 | 6 | 0
  10-1074 (Day- 14) |  |  | 289.86 [207.92 to 311.78] |
  10-1074 (Day- 28): number analyzed (Participants) | 0 | 0 | 5 | 0
  10-1074 (Day- 28) |  |  | 242.22 [140.97 to 253.34] |
  10-1074 (Day- 56): number analyzed (Participants) | 0 | 0 | 5 | 0
  10-1074 (Day- 56) |  |  | 98.27 [29.65 to 124.97] |
  10-1074 (Day-112): number analyzed (Participants) | 0 | 0 | 5 | 0
  10-1074 (Day-112) |  |  | 23.96 [8.04 to 26.39] |
  10-1074 (Day-168): number analyzed (Participants) | 0 | 0 | 4 | 0
  10-1074 (Day-168) |  |  | 8.60 [6.27 to 11.17] |
  10-1074 (Day-224): number analyzed (Participants) | 0 | 0 | 0 | 0
  10-1074 (Day-280): number analyzed (Participants) | 0 | 0 | 4 | 0
  10-1074 (Day-280) |  |  | 0.59 [0.21 to 2.11] |
  10-1074 (Day-336): number analyzed (Participants) | 0 | 0 | 2 | 0
  10-1074 (Day-336) |  |  | 2.44 [1.32 to 3.55] |
  PGDM1400 (Day- 0): number analyzed (Participants) | 0 | 6 | 0 | 9
  PGDM1400 (Day- 0) |  | 0.02 [0.02 to 0.02] |  | 0.02 [0.02 to 0.02]
  PGDM1400 (Day- 3): number analyzed (Participants) | 0 | 6 | 0 | 9
  PGDM1400 (Day- 3) |  | 251.54 [234.47 to 273.48] |  | 231.33 [203.73 to 319.27]
  PGDM1400 (Day- 6): number analyzed (Participants) | 0 | 6 | 0 | 9
  PGDM1400 (Day- 6) |  | 182.23 [160.51 to 186.36] |  | 173.81 [168.63 to 177.65]
  PGDM1400 (Day- 14): number analyzed (Participants) | 0 | 6 | 0 | 9
  PGDM1400 (Day- 14) |  | 139.77 [134.94 to 146.76] |  | 126.56 [113.27 to 146.69]
  PGDM1400 (Day- 28): number analyzed (Participants) | 0 | 6 | 0 | 9
  PGDM1400 (Day- 28) |  | 70.92 [67.17 to 73.87] |  | 71.60 [52.74 to 77.35]
  PGDM1400 (Day- 56): number analyzed (Participants) | 0 | 6 | 0 | 9
  PGDM1400 (Day- 56) |  | 27.88 [26.68 to 31.56] |  | 33.70 [19.33 to 39.98]
  PGDM1400 (Day- 84): number analyzed (Participants) | 0 | 0 | 0 | 9
  PGDM1400 (Day- 84) |  |  |  | 12.26 [7.20 to 15.87]
  PGDM1400 (Day-112): number analyzed (Participants) | 0 | 5 | 0 | 6
  PGDM1400 (Day-112) |  | 5.50 [4.63 to 6.04] |  | 4.99 [3.81 to 7.11]
  PGDM1400 (Day-140): number analyzed (Participants) | 0 | 0 | 0 | 3
  PGDM1400 (Day-140) |  |  |  | 3.49 [2.34 to 24.78]
  PGDM1400 (Day-168): number analyzed (Participants) | 0 | 4 | 0 | 2
  PGDM1400 (Day-168) |  | 1.08 [1.02 to 1.10] |  | 1.51 [1.14 to 1.88]
  PGDM1400 (Day-224): number analyzed (Participants) | 0 | 1 | 0 | 5
  PGDM1400 (Day-224) |  | 0.26 [0.26 to 0.26] |  | 2.21 [0.88 to 6.24]
  PGDM1400 (Day-280): number analyzed (Participants) | 0 | 1 | 0 | 7
  PGDM1400 (Day-280) |  | 0.09 [0.09 to 0.09] |  | 0.50 [0.23 to 1.41]
  PGDM1400 (Day-336): number analyzed (Participants) | 0 | 2 | 0 | 8
  PGDM1400 (Day-336) |  | 0.02 [0.02 to 0.02] |  | 0.25 [0.08 to 0.65]
  PGDM1400 (Day-392): number analyzed (Participants) | 0 | 0 | 0 | 7
  PGDM1400 (Day-392) |  |  |  | 0.04 [0.02 to 0.11]
  PGDM1400 (Day-448): number analyzed (Participants) | 0 | 0 | 0 | 7
  PGDM1400 (Day-448) |  |  |  | 0.02 [0.02 to 0.03]
  PGT121 (Day- 0): number analyzed (Participants) | 6 | 0 | 0 | 9
  PGT121 (Day- 0) | 0.05 [0.05 to 0.05] |  |  | 0.05 [0.05 to 0.05]
  PGT121 (Day- 3): number analyzed (Participants) | 6 | 0 | 0 | 9
  PGT121 (Day- 3) | 196.57 [172.85 to 210.31] |  |  | 181.38 [157.86 to 219.10]
  PGT121 (Day- 6): number analyzed (Participants) | 6 | 0 | 0 | 9
  PGT121 (Day- 6) | 129.35 [116.95 to 137.34] |  |  | 130.98 [128.10 to 137.61]
  PGT121 (Day- 14): number analyzed (Participants) | 6 | 0 | 0 | 9
  PGT121 (Day- 14) | 80.12 [79.07 to 86.22] |  |  | 90.47 [84.84 to 100.59]
  PGT121 (Day- 28): number analyzed (Participants) | 6 | 0 | 0 | 9
  PGT121 (Day- 28) | 44.46 [40.81 to 50.03] |  |  | 56.75 [45.47 to 64.49]
  PGT121 (Day- 56): number analyzed (Participants) | 6 | 0 | 0 | 9
  PGT121 (Day- 56) | 22.08 [18.83 to 23.24] |  |  | 29.32 [19.33 to 31.85]
  PGT121 (Day- 84): number analyzed (Participants) | 0 | 0 | 0 | 9
  PGT121 (Day- 84) |  |  |  | 15.00 [8.83 to 16.35]
  PGT121 (Day-112): number analyzed (Participants) | 6 | 0 | 0 | 6
  PGT121 (Day-112) | 4.03 [3.45 to 5.97] |  |  | 5.82 [5.60 to 10.02]
  PGT121 (Day-140): number analyzed (Participants) | 0 | 0 | 0 | 3
  PGT121 (Day-140) |  |  |  | 6.08 [4.06 to 27.62]
  PGT121 (Day-168): number analyzed (Participants) | 4 | 0 | 0 | 2
  PGT121 (Day-168) | 1.70 [0.88 to 3.28] |  |  | 2.72 [2.02 to 3.41]
  PGT121 (Day-224): number analyzed (Participants) | 1 | 0 | 0 | 5
  PGT121 (Day-224) | 0.31 [0.31 to 0.31] |  |  | 4.16 [2.08 to 11.28]
  PGT121 (Day-280): number analyzed (Participants) | 0 | 0 | 0 | 7
  PGT121 (Day-280) |  |  |  | 1.46 [0.74 to 3.46]
  PGT121 (Day-336): number analyzed (Participants) | 5 | 0 | 0 | 8
  PGT121 (Day-336) | 0.05 [0.05 to 0.11] |  |  | 0.71 [0.34 to 1.43]
  PGT121 (Day-392): number analyzed (Participants) | 0 | 0 | 0 | 7
  PGT121 (Day-392) |  |  |  | 0.18 [0.14 to 0.49]
  PGT121 (Day-448): number analyzed (Participants) | 0 | 0 | 0 | 7
  PGT121 (Day-448) |  |  |  | 0.05 [0.05 to 0.19]
  VRC07-523LS (Day- 0) | 0.01 [0.01 to 0.02] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.01]
  VRC07-523LS (Day- 3) | 265.97 [262.58 to 300.62] | 239.32 [224.13 to 264.34] | 173.73 [145.91 to 186.22] | 230.06 [199.85 to 333.96]
  VRC07-523LS (Day- 6) | 171.02 [158.01 to 209.24] | 176.51 [158.50 to 183.85] | 171.62 [164.76 to 176.61] | 169.54 [155.85 to 182.30]
  VRC07-523LS (Day- 14) | 134.44 [128.24 to 135.66] | 139.18 [105.71 to 155.86] | 105.05 [85.34 to 138.74] | 133.03 [120.16 to 146.62]
  VRC07-523LS (Day- 28): number analyzed (Participants) | 6 | 6 | 5 | 9
  VRC07-523LS (Day- 28) | 94.58 [88.61 to 102.26] | 96.17 [83.80 to 110.65] | 87.91 [85.13 to 96.66] | 96.52 [94.26 to 104.18]
  VRC07-523LS (Day- 56): number analyzed (Participants) | 6 | 6 | 5 | 9
  VRC07-523LS (Day- 56) | 60.53 [55.78 to 62.70] | 56.91 [56.03 to 58.35] | 56.91 [34.69 to 61.74] | 60.24 [53.64 to 67.05]
  VRC07-523LS (Day- 84): number analyzed (Participants) | 0 | 0 | 0 | 9
  VRC07-523LS (Day- 84) |  |  |  | 41.64 [31.11 to 44.37]
  VRC07-523LS (Day-112): number analyzed (Participants) | 6 | 5 | 5 | 6
  VRC07-523LS (Day-112) | 24.93 [20.69 to 26.88] | 31.65 [20.09 to 33.07] | 28.18 [11.53 to 30.55] | 26.07 [19.85 to 33.70]
  VRC07-523LS (Day-140): number analyzed (Participants) | 0 | 0 | 0 | 3
  VRC07-523LS (Day-140) |  |  |  | 13.94 [13.09 to 44.99]
  VRC07-523LS (Day-168): number analyzed (Participants) | 4 | 4 | 4 | 2
  VRC07-523LS (Day-168) | 14.45 [12.37 to 16.66] | 12.57 [10.74 to 14.17] | 11.57 [9.73 to 12.35] | 9.98 [9.46 to 10.50]
  VRC07-523LS (Day-224): number analyzed (Participants) | 1 | 1 | 0 | 5
  VRC07-523LS (Day-224) | 8.47 [8.47 to 8.47] | 11.24 [11.24 to 11.24] |  | 22.66 [5.51 to 39.86]
  VRC07-523LS (Day-280): number analyzed (Participants) | 0 | 1 | 4 | 7
  VRC07-523LS (Day-280) |  | 3.88 [3.88 to 3.88] | 1.81 [0.34 to 3.33] | 14.85 [5.99 to 15.82]
  VRC07-523LS (Day-336): number analyzed (Participants) | 5 | 2 | 3 | 8
  VRC07-523LS (Day-336) | 1.33 [1.08 to 1.38] | 1.31 [1.16 to 1.46] | 1.48 [0.85 to 2.34] | 7.49 [4.31 to 10.51]
  VRC07-523LS (Day-392): number analyzed (Participants) | 0 | 0 | 0 | 7
  VRC07-523LS (Day-392) |  |  |  | 2.73 [1.75 to 5.00]
  VRC07-523LS (Day-448): number analyzed (Participants) | 0 | 0 | 0 | 7
  VRC07-523LS (Day-448) |  |  |  | 1.10 [0.69 to 2.37]

14. Secondary Outcome: Magnitudes of TZM-bl Cells Responses Against a Panel of Env Pseudotyped Viruses for All Participants
Description: as for outcome 12
Time Frame: Measured during Screening, Days 0, 3, 28, 56, 112, 140*, 168*, 224* Days with * are only available for T4
Population: All participants enrolled with available neutralizing antibody data. Visits with 0 participants are due to: (1) Isolates were mAb-specific and only assayed for the treatment arms that received the specific mAbs. (2) Treatment group T4 had more scheduled sample collection visits than treatment groups T1-T3.
Measure: Median (Inter-Quartile Range); unit: Relative luminescence units (RLU)
Arm/Group | T1: PGT121 + VRC07-523LS mo 0 | T2: PGDM1400 + VRC07-523LS mo 0 | T3: 10-1074 + VRC07-523LS | T4: PGT121 + PGDM1400 + VRC07-523LS mo(0, 4)
Number analyzed (Participants) | 6 | 6 | 6 | 9
Relative luminescence units (RLU)
  6540.v4.c1 (Day- 0): number analyzed (Participants) | 0 | 0 | 0 | 9
  6540.v4.c1 (Day- 0) |  |  |  | 5.00 [5.00 to 5.00]
  6540.v4.c1 (Day- 3): number analyzed (Participants) | 0 | 0 | 0 | 9
  6540.v4.c1 (Day- 3) |  |  |  | 13187.62 [9441.20 to 18617.3]
  6540.v4.c1 (Day- 28): number analyzed (Participants) | 0 | 0 | 0 | 9
  6540.v4.c1 (Day- 28) |  |  |  | 2083.51 [1820.80 to 2758.25]
  6540.v4.c1 (Day- 56): number analyzed (Participants) | 0 | 0 | 0 | 9
  6540.v4.c1 (Day- 56) |  |  |  | 774.27 [530.97 to 919.39]
  6540.v4.c1 (Day-112): number analyzed (Participants) | 0 | 0 | 0 | 6
  6540.v4.c1 (Day-112) |  |  |  | 82.11 [61.03 to 98.13]
  6540.v4.c1 (Day-140): number analyzed (Participants) | 0 | 0 | 0 | 3
  6540.v4.c1 (Day-140) |  |  |  | 45.07 [25.03 to 650.34]
  6540.v4.c1 (Day-168): number analyzed (Participants) | 0 | 0 | 0 | 2
  6540.v4.c1 (Day-168) |  |  |  | 14.74 [9.87 to 19.62]
  6540.v4.c1 (Day-224): number analyzed (Participants) | 0 | 0 | 0 | 5
  6540.v4.c1 (Day-224) |  |  |  | 27.66 [5.00 to 64.76]
  CH505TF.N334S.N160A.N280D.1 (Day- 0): number analyzed (Participants) | 0 | 0 | 0 | 9
  CH505TF.N334S.N160A.N280D.1 (Day- 0) |  |  |  | 5.00 [5.00 to 5.00]
  CH505TF.N334S.N160A.N280D.1 (Day- 3): number analyzed (Participants) | 0 | 0 | 0 | 9
  CH505TF.N334S.N160A.N280D.1 (Day- 3) |  |  |  | 13343.35 [9088.55 to 18308.4]
  CH505TF.N334S.N160A.N280D.1 (Day- 28): number analyzed (Participants) | 0 | 0 | 0 | 9
  CH505TF.N334S.N160A.N280D.1 (Day- 28) |  |  |  | 3000.56 [2917.48 to 3828.38]
  CH505TF.N334S.N160A.N280D.1 (Day- 56): number analyzed (Participants) | 0 | 0 | 0 | 9
  CH505TF.N334S.N160A.N280D.1 (Day- 56) |  |  |  | 1751.70 [1019.21 to 1968.06]
  CH505TF.N334S.N160A.N280D.1 (Day-112): number analyzed (Participants) | 0 | 0 | 0 | 6
  CH505TF.N334S.N160A.N280D.1 (Day-112) |  |  |  | 339.83 [296.59 to 554.03]
  CH505TF.N334S.N160A.N280D.1 (Day-140): number analyzed (Participants) | 0 | 0 | 0 | 3
  CH505TF.N334S.N160A.N280D.1 (Day-140) |  |  |  | 270.10 [176.30 to 1416.59]
  CH505TF.N334S.N160A.N280D.1 (Day-168): number analyzed (Participants) | 0 | 0 | 0 | 2
  CH505TF.N334S.N160A.N280D.1 (Day-168) |  |  |  | 111.35 [86.07 to 136.63]
  CH505TF.N334S.N160A.N280D.1 (Day-224): number analyzed (Participants) | 0 | 0 | 0 | 5
  CH505TF.N334S.N160A.N280D.1 (Day-224) |  |  |  | 206.62 [105.46 to 429.44]
  CNE55.N160K (Day- 0) | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  CNE55.N160K (Day- 3) | 917.25 [686.59 to 1286.70] | 816.88 [725.91 to 847.67] | 438.49 [357.53 to 535.46] | 466.43 [421.07 to 1000.34]
  CNE55.N160K (Day- 28): number analyzed (Participants) | 6 | 6 | 5 | 9
  CNE55.N160K (Day- 28) | 259.58 [212.45 to 323.50] | 188.55 [161.50 to 208.80] | 206.12 [171.05 to 268.36] | 158.46 [146.09 to 233.05]
  CNE55.N160K (Day- 56): number analyzed (Participants) | 6 | 6 | 5 | 9
  CNE55.N160K (Day- 56) | 105.02 [91.83 to 118.53] | 91.57 [80.40 to 117.12] | 152.21 [95.36 to 188.88] | 131.95 [98.57 to 134.34]
  CNE55.N160K (Day-112): number analyzed (Participants) | 6 | 5 | 5 | 6
  CNE55.N160K (Day-112) | 28.65 [25.10 to 36.11] | 10.00 [10.00 to 20.95] | 47.58 [10.00 to 59.38] | 47.57 [30.49 to 65.17]
  CNE55.N160K (Day-140): number analyzed (Participants) | 0 | 0 | 0 | 3
  CNE55.N160K (Day-140) |  |  |  | 18.76 [17.13 to 55.76]
  CNE55.N160K (Day-168): number analyzed (Participants) | 0 | 0 | 0 | 2
  CNE55.N160K (Day-168) |  |  |  | 13.27 [9.14 to 17.41]
  CNE55.N160K (Day-224): number analyzed (Participants) | 0 | 0 | 0 | 5
  CNE55.N160K (Day-224) |  |  |  | 37.80 [14.65 to 58.52]
  T250-4 (Day- 0): number analyzed (Participants) | 6 | 6 | 6 | 0
  T250-4 (Day- 0) | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] |
  T250-4 (Day- 3): number analyzed (Participants) | 6 | 6 | 6 | 0
  T250-4 (Day- 3) | 32029.39 [28181.95 to 41032.5] | 91301.02 [79640.01 to 114904.] | 35379.15 [25190.07 to 44080.8] |
  T250-4 (Day- 28): number analyzed (Participants) | 6 | 6 | 5 | 0
  T250-4 (Day- 28) | 6458.16 [5518.54 to 7452.56] | 27318.99 [23401.71 to 30312.3] | 13028.85 [11586.88 to 14345.8] |
  T250-4 (Day- 56): number analyzed (Participants) | 6 | 6 | 5 | 0
  T250-4 (Day- 56) | 2016.84 [1800.34 to 2646.68] | 7523.58 [6020.17 to 8716.04] | 6515.27 [2851.83 to 7625.68] |
  T250-4 (Day-112): number analyzed (Participants) | 6 | 5 | 5 | 0
  T250-4 (Day-112) | 300.37 [266.45 to 650.96] | 800.00 [618.17 to 837.77] | 928.27 [529.97 to 1449.78] |

15. Secondary Outcome: Magnitude of Neutralizing Activity Against a Panel of Env Pseudotyped Reference Viruses in TZM-bl Cells for All Participants
Description: as for outcome 12
Time Frame: Measured during Screening, Days 0*, 3, 28, 56*, 112, 140*, 224* Days with * are only available for T4
Population: All participants enrolled with available neutralizing antibody data. Visits with 0 participants are due to: Treatment group T4 had more scheduled sample collection visits than treatment groups T1-T3.
Measure: Median (Inter-Quartile Range); unit: Relative luminescence units (RLU)
Arm/Group | T1: PGT121 + VRC07-523LS mo 0 | T2: PGDM1400 + VRC07-523LS mo 0 | T3: 10-1074 + VRC07-523LS | T4: PGT121 + PGDM1400 + VRC07-523LS mo(0, 4)
Number analyzed (Participants) | 6 | 6 | 6 | 9
Relative luminescence units (RLU)
  0330.v4.c3 (Day- 0): number analyzed (Participants) | 0 | 0 | 0 | 9
  0330.v4.c3 (Day- 0) |  |  |  | 5.00 [5.00 to 5.00]
  0330.v4.c3 (Day- 3) | 6396.28 [6080.23 to 6735.71] | 74297.85 [52044.99 to 88109.3] | 6121.19 [3340.46 to 12217.9] | 89412.79 [81404.07 to 133261.]
  0330.v4.c3 (Day- 28): number analyzed (Participants) | 6 | 6 | 5 | 9
  0330.v4.c3 (Day- 28) | 1714.47 [1464.17 to 1902.42] | 12264.66 [10502.90 to 16471.8] | 1117.61 [1052.55 to 1387.42] | 19794.60 [12324.14 to 23999.2]
  0330.v4.c3 (Day- 56): number analyzed (Participants) | 0 | 0 | 0 | 9
  0330.v4.c3 (Day- 56) |  |  |  | 5217.82 [3172.08 to 6238.47]
  0330.v4.c3 (Day-112): number analyzed (Participants) | 6 | 5 | 5 | 6
  0330.v4.c3 (Day-112) | 242.94 [181.50 to 300.77] | 1216.32 [807.32 to 1581.69] | 209.33 [99.69 to 222.71] | 611.93 [453.02 to 750.19]
  0330.v4.c3 (Day-140): number analyzed (Participants) | 0 | 0 | 0 | 3
  0330.v4.c3 (Day-140) |  |  |  | 589.67 [389.86 to 3617.62]
  0330.v4.c3 (Day-224): number analyzed (Participants) | 0 | 0 | 0 | 5
  0330.v4.c3 (Day-224) |  |  |  | 343.14 [116.53 to 669.99]
  3426.v5.c17 (Day- 0): number analyzed (Participants) | 0 | 0 | 0 | 9
  3426.v5.c17 (Day- 0) |  |  |  | 5.00 [5.00 to 5.00]
  3426.v5.c17 (Day- 3) | 16924.30 [14561.42 to 20967.7] | 144218.5 [93034.17 to 406283.] | 9665.13 [7360.48 to 11861.0] | 368712.2 [259743.1 to 390143.]
  3426.v5.c17 (Day- 28): number analyzed (Participants) | 6 | 6 | 5 | 9
  3426.v5.c17 (Day- 28) | 3041.45 [2966.23 to 3290.51] | 32852.84 [26522.32 to 46738.8] | 2676.34 [2001.12 to 2816.62] | 66390.30 [64990.87 to 97262.7]
  3426.v5.c17 (Day- 56): number analyzed (Participants) | 0 | 0 | 0 | 9
  3426.v5.c17 (Day- 56) |  |  |  | 24227.08 [8980.36 to 33004.1]
  3426.v5.c17 (Day-112): number analyzed (Participants) | 6 | 5 | 5 | 6
  3426.v5.c17 (Day-112) | 362.56 [274.34 to 473.09] | 1488.31 [993.10 to 1671.42] | 447.09 [97.17 to 463.62] | 1288.16 [1082.09 to 2303.78]
  3426.v5.c17 (Day-140): number analyzed (Participants) | 0 | 0 | 0 | 3
  3426.v5.c17 (Day-140) |  |  |  | 822.84 [540.23 to 14854.5]
  3426.v5.c17 (Day-224): number analyzed (Participants) | 0 | 0 | 0 | 5
  3426.v5.c17 (Day-224) |  |  |  | 537.48 [182.83 to 1909.54]
  377.v4.c09 (Day- 0): number analyzed (Participants) | 0 | 0 | 0 | 9
  377.v4.c09 (Day- 0) |  |  |  | 5.00 [5.00 to 5.00]
  377.v4.c09 (Day- 3) | 441.18 [411.01 to 504.06] | 255.40 [209.29 to 281.66] | 380.32 [278.05 to 459.21] | 591.58 [482.75 to 800.29]
  377.v4.c09 (Day- 28): number analyzed (Participants) | 6 | 6 | 5 | 9
  377.v4.c09 (Day- 28) | 108.14 [102.75 to 114.54] | 63.14 [58.58 to 72.02] | 116.45 [96.92 to 117.19] | 179.21 [127.50 to 211.82]
  377.v4.c09 (Day- 56): number analyzed (Participants) | 0 | 0 | 0 | 9
  377.v4.c09 (Day- 56) |  |  |  | 85.74 [59.71 to 97.87]
  377.v4.c09 (Day-112): number analyzed (Participants) | 6 | 5 | 5 | 6
  377.v4.c09 (Day-112) | 16.27 [12.25 to 18.09] | 5.00 [5.00 to 5.00] | 14.68 [5.00 to 15.14] | 17.94 [13.93 to 26.97]
  377.v4.c09 (Day-140): number analyzed (Participants) | 0 | 0 | 0 | 3
  377.v4.c09 (Day-140) |  |  |  | 14.48 [9.74 to 91.02]
  377.v4.c09 (Day-224): number analyzed (Participants) | 0 | 0 | 0 | 5
  377.v4.c09 (Day-224) |  |  |  | 17.09 [5.00 to 37.52]
  AC10.0.29 (Day- 0): number analyzed (Participants) | 0 | 0 | 0 | 9
  AC10.0.29 (Day- 0) |  |  |  | 5.00 [5.00 to 5.00]
  AC10.0.29 (Day- 3) | 3307.09 [3201.01 to 3589.36] | 1198.26 [1097.26 to 1305.86] | 2763.45 [2425.04 to 3413.11] | 3854.76 [3252.76 to 5347.95]
  AC10.0.29 (Day- 28): number analyzed (Participants) | 6 | 6 | 5 | 9
  AC10.0.29 (Day- 28) | 730.53 [710.40 to 751.62] | 285.36 [277.39 to 333.60] | 842.99 [802.47 to 1038.29] | 1039.01 [761.35 to 1117.14]
  AC10.0.29 (Day- 56): number analyzed (Participants) | 0 | 0 | 0 | 9
  AC10.0.29 (Day- 56) |  |  |  | 500.07 [312.83 to 597.44]
  AC10.0.29 (Day-112): number analyzed (Participants) | 6 | 5 | 5 | 6
  AC10.0.29 (Day-112) | 58.82 [50.35 to 97.12] | 37.55 [34.74 to 44.08] | 152.58 [28.49 to 154.06] | 85.57 [59.92 to 153.51]
  AC10.0.29 (Day-140): number analyzed (Participants) | 0 | 0 | 0 | 3
  AC10.0.29 (Day-140) |  |  |  | 75.66 [51.59 to 455.20]
  AC10.0.29 (Day-224): number analyzed (Participants) | 0 | 0 | 0 | 5
  AC10.0.29 (Day-224) |  |  |  | 57.51 [22.44 to 162.14]
  Ce1176_A3 (Day- 0): number analyzed (Participants) | 0 | 0 | 0 | 9
  Ce1176_A3 (Day- 0) |  |  |  | 5.00 [5.00 to 5.00]
  Ce1176_A3 (Day- 3) | 11645.78 [9518.45 to 12116.3] | 537.29 [459.87 to 586.96] | 4781.11 [3229.13 to 7086.33] | 8628.18 [6578.27 to 12370.5]
  Ce1176_A3 (Day- 28): number analyzed (Participants) | 6 | 6 | 5 | 9
  Ce1176_A3 (Day- 28) | 1869.57 [1853.02 to 2232.85] | 137.78 [109.83 to 145.47] | 1475.03 [954.07 to 1488.48] | 2081.67 [1688.46 to 2313.62]
  Ce1176_A3 (Day- 56): number analyzed (Participants) | 0 | 0 | 0 | 9
  Ce1176_A3 (Day- 56) |  |  |  | 842.00 [564.10 to 1444.53]
  Ce1176_A3 (Day-112): number analyzed (Participants) | 6 | 5 | 5 | 6
  Ce1176_A3 (Day-112) | 139.63 [95.90 to 265.94] | 28.13 [17.77 to 28.27] | 165.45 [41.81 to 206.47] | 199.63 [160.77 to 372.51]
  Ce1176_A3 (Day-140): number analyzed (Participants) | 0 | 0 | 0 | 3
  Ce1176_A3 (Day-140) |  |  |  | 205.80 [128.04 to 963.06]
  Ce1176_A3 (Day-224): number analyzed (Participants) | 0 | 0 | 0 | 5
  Ce1176_A3 (Day-224) |  |  |  | 101.07 [48.45 to 381.19]
  DU156.12 (Day- 0): number analyzed (Participants) | 0 | 0 | 0 | 9
  DU156.12 (Day- 0) |  |  |  | 5.00 [5.00 to 5.00]
  DU156.12 (Day- 3) | 18539.26 [17172.56 to 23579.6] | 27452.85 [26185.95 to 28715.5] | 10841.11 [5764.85 to 14232.2] | 84807.92 [32946.35 to 107084.]
  DU156.12 (Day- 28): number analyzed (Participants) | 6 | 6 | 5 | 9
  DU156.12 (Day- 28) | 4812.81 [4150.62 to 5672.03] | 6655.88 [5796.38 to 6937.67] | 2989.42 [2466.94 to 3703.45] | 14630.79 [12167.11 to 23357.8]
  DU156.12 (Day- 56): number analyzed (Participants) | 0 | 0 | 0 | 9
  DU156.12 (Day- 56) |  |  |  | 3915.57 [2878.16 to 5887.10]
  DU156.12 (Day-112): number analyzed (Participants) | 6 | 5 | 5 | 6
  DU156.12 (Day-112) | 632.13 [498.04 to 735.92] | 620.22 [503.29 to 741.76] | 629.27 [199.42 to 648.10] | 744.96 [605.25 to 1202.94]
  DU156.12 (Day-140): number analyzed (Participants) | 0 | 0 | 0 | 3
  DU156.12 (Day-140) |  |  |  | 627.31 [437.57 to 4019.46]
  DU156.12 (Day-224): number analyzed (Participants) | 0 | 0 | 0 | 5
  DU156.12 (Day-224) |  |  |  | 578.62 [161.72 to 832.75]
  DU172.17 (Day- 0): number analyzed (Participants) | 0 | 0 | 0 | 9
  DU172.17 (Day- 0) |  |  |  | 5.00 [5.00 to 5.00]
  DU172.17 (Day- 3) | 1518.88 [1163.34 to 1850.98] | 448.77 [342.15 to 495.87] | 1315.85 [1037.49 to 1898.68] | 1631.83 [1393.41 to 1944.91]
  DU172.17 (Day- 28): number analyzed (Participants) | 6 | 6 | 5 | 9
  DU172.17 (Day- 28) | 434.85 [402.56 to 448.27] | 170.68 [119.08 to 194.91] | 398.72 [383.47 to 448.60] | 413.93 [332.95 to 532.05]
  DU172.17 (Day- 56): number analyzed (Participants) | 0 | 0 | 0 | 9
  DU172.17 (Day- 56) |  |  |  | 187.19 [162.90 to 224.12]
  DU172.17 (Day-112): number analyzed (Participants) | 6 | 5 | 5 | 6
  DU172.17 (Day-112) | 45.10 [37.03 to 71.39] | 16.67 [5.00 to 22.47] | 61.30 [16.72 to 66.06] | 56.99 [46.08 to 78.16]
  DU172.17 (Day-140): number analyzed (Participants) | 0 | 0 | 0 | 3
  DU172.17 (Day-140) |  |  |  | 43.33 [27.32 to 178.56]
  DU172.17 (Day-224): number analyzed (Participants) | 0 | 0 | 0 | 5
  DU172.17 (Day-224) |  |  |  | 33.71 [11.22 to 72.76]
  PVO.4 (Day- 0): number analyzed (Participants) | 0 | 0 | 0 | 9
  PVO.4 (Day- 0) |  |  |  | 5.00 [5.00 to 5.00]
  PVO.4 (Day- 3) | 1834.12 [1630.50 to 2102.57] | 773.42 [697.14 to 903.36] | 1918.35 [1098.33 to 2093.31] | 2078.34 [1885.71 to 2315.32]
  PVO.4 (Day- 28): number analyzed (Participants) | 6 | 6 | 5 | 9
  PVO.4 (Day- 28) | 523.42 [443.00 to 527.84] | 244.89 [240.35 to 248.11] | 548.04 [529.82 to 634.73] | 611.64 [557.45 to 649.11]
  PVO.4 (Day- 56): number analyzed (Participants) | 0 | 0 | 0 | 9
  PVO.4 (Day- 56) |  |  |  | 316.00 [215.71 to 363.56]
  PVO.4 (Day-112): number analyzed (Participants) | 6 | 5 | 5 | 6
  PVO.4 (Day-112) | 80.37 [67.76 to 93.09] | 50.58 [46.64 to 54.40] | 99.15 [40.87 to 104.77] | 92.98 [76.81 to 112.41]
  PVO.4 (Day-140): number analyzed (Participants) | 0 | 0 | 0 | 3
  PVO.4 (Day-140) |  |  |  | 45.61 [40.70 to 230.18]
  PVO.4 (Day-224): number analyzed (Participants) | 0 | 0 | 0 | 5
  PVO.4 (Day-224) |  |  |  | 58.33 [20.52 to 110.43]
  RHPA4259.7 (Day- 0): number analyzed (Participants) | 0 | 0 | 0 | 9
  RHPA4259.7 (Day- 0) |  |  |  | 5.00 [5.00 to 5.00]
  RHPA4259.7 (Day- 3) | 15786.94 [13562.87 to 19915.2] | 4313.94 [3709.44 to 5821.77] | 6847.08 [5023.53 to 9267.51] | 11323.55 [10578.46 to 15367.3]
  RHPA4259.7 (Day- 28): number analyzed (Participants) | 6 | 6 | 5 | 9
  RHPA4259.7 (Day- 28) | 3718.80 [3383.58 to 4228.20] | 1748.53 [1639.88 to 1788.12] | 2996.20 [2164.60 to 3266.73] | 3560.23 [3338.05 to 3839.56]
  RHPA4259.7 (Day- 56): number analyzed (Participants) | 0 | 0 | 0 | 9
  RHPA4259.7 (Day- 56) |  |  |  | 2114.58 [1601.57 to 2685.28]
  RHPA4259.7 (Day-112): number analyzed (Participants) | 6 | 5 | 5 | 6
  RHPA4259.7 (Day-112) | 663.30 [477.36 to 857.77] | 506.64 [364.10 to 511.53] | 528.88 [267.50 to 555.36] | 562.77 [485.83 to 788.27]
  RHPA4259.7 (Day-140): number analyzed (Participants) | 0 | 0 | 0 | 3
  RHPA4259.7 (Day-140) |  |  |  | 384.75 [279.01 to 1524.80]
  RHPA4259.7 (Day-224): number analyzed (Participants) | 0 | 0 | 0 | 5
  RHPA4259.7 (Day-224) |  |  |  | 406.26 [131.41 to 768.36]
  SC422661.8 (Day- 0): number analyzed (Participants) | 0 | 0 | 0 | 9
  SC422661.8 (Day- 0) |  |  |  | 5.00 [5.00 to 5.00]
  SC422661.8 (Day- 3) | 3925.17 [3766.76 to 4704.83] | 2519.42 [1997.20 to 2761.47] | 3601.22 [2513.76 to 4602.54] | 5345.96 [3397.00 to 5947.47]
  SC422661.8 (Day- 28): number analyzed (Participants) | 6 | 6 | 5 | 9
  SC422661.8 (Day- 28) | 1389.90 [1302.50 to 1530.08] | 1035.29 [725.16 to 1287.34] | 1408.81 [1227.23 to 1411.60] | 1377.52 [1147.39 to 1725.51]
  SC422661.8 (Day- 56): number analyzed (Participants) | 0 | 0 | 0 | 9
  SC422661.8 (Day- 56) |  |  |  | 765.08 [625.41 to 991.03]
  SC422661.8 (Day-112): number analyzed (Participants) | 6 | 5 | 5 | 6
  SC422661.8 (Day-112) | 213.39 [186.07 to 275.41] | 163.39 [156.87 to 174.58] | 219.98 [95.53 to 267.65] | 189.00 [183.79 to 276.06]
  SC422661.8 (Day-140): number analyzed (Participants) | 0 | 0 | 0 | 3
  SC422661.8 (Day-140) |  |  |  | 120.06 [103.68 to 514.08]
  SC422661.8 (Day-224): number analyzed (Participants) | 0 | 0 | 0 | 5
  SC422661.8 (Day-224) |  |  |  | 192.58 [53.76 to 269.09]
  T263-8 (Day- 0): number analyzed (Participants) | 0 | 0 | 0 | 9
  T263-8 (Day- 0) |  |  |  | 5.00 [5.00 to 5.00]
  T263-8 (Day- 3) | 2776.59 [2281.26 to 3281.31] | 8794.97 [8451.76 to 11791.8] | 1811.12 [1236.81 to 1988.47] | 10506.56 [7759.25 to 12494.5]
  T263-8 (Day- 28): number analyzed (Participants) | 6 | 6 | 5 | 9
  T263-8 (Day- 28) | 652.72 [623.52 to 799.07] | 2180.36 [2077.13 to 2332.70] | 709.37 [659.45 to 713.01] | 2076.06 [2000.37 to 2452.00]
  T263-8 (Day- 56): number analyzed (Participants) | 0 | 0 | 0 | 9
  T263-8 (Day- 56) |  |  |  | 789.69 [562.19 to 1124.91]
  T263-8 (Day-112): number analyzed (Participants) | 6 | 5 | 5 | 6
  T263-8 (Day-112) | 168.55 [139.98 to 176.97] | 260.69 [204.99 to 326.59] | 156.80 [77.23 to 174.38] | 169.57 [128.05 to 260.28]
  T263-8 (Day-140): number analyzed (Participants) | 0 | 0 | 0 | 3
  T263-8 (Day-140) |  |  |  | 99.18 [83.78 to 680.21]
  T263-8 (Day-224): number analyzed (Participants) | 0 | 0 | 0 | 5
  T263-8 (Day-224) |  |  |  | 130.83 [36.33 to 281.58]
  TRO.11 (Day- 0): number analyzed (Participants) | 0 | 0 | 0 | 9
  TRO.11 (Day- 0) |  |  |  | 5.00 [5.00 to 5.00]
  TRO.11 (Day- 3) | 7813.45 [7044.18 to 8400.16] | 887.77 [744.43 to 1025.75] | 4253.82 [2683.78 to 5150.14] | 8880.74 [6305.55 to 9378.98]
  TRO.11 (Day- 28): number analyzed (Participants) | 6 | 6 | 5 | 9
  TRO.11 (Day- 28) | 1503.04 [1409.62 to 1726.44] | 249.19 [202.44 to 318.67] | 1085.04 [954.52 to 1375.31] | 1963.86 [1656.59 to 2787.73]
  TRO.11 (Day- 56): number analyzed (Participants) | 0 | 0 | 0 | 9
  TRO.11 (Day- 56) |  |  |  | 1023.42 [611.40 to 1196.50]
  TRO.11 (Day-112): number analyzed (Participants) | 6 | 5 | 5 | 6
  TRO.11 (Day-112) | 116.90 [101.82 to 156.21] | 73.93 [37.19 to 75.09] | 193.46 [66.49 to 206.92] | 182.49 [153.74 to 287.64]
  TRO.11 (Day-140): number analyzed (Participants) | 0 | 0 | 0 | 3
  TRO.11 (Day-140) |  |  |  | 146.55 [95.84 to 783.56]
  TRO.11 (Day-224): number analyzed (Participants) | 0 | 0 | 0 | 5
  TRO.11 (Day-224) |  |  |  | 111.00 [47.82 to 333.09]

ADVERSE EVENTS:
Time Frame: The study Unsolicited AE reporting time frame is from study enrollment of a trial participant to (and including) Day 336 for T1-T3 and Day 448 for T4. The Solicited AE assessment were collected through 3 full days after each vaccination (vaccinations were given at Day 0 for T1-T4 and Day 112 for T4).
Arm/Group | T1: PGT121 + VRC07-523LS mo 0 | T2: PGDM1400 + VRC07-523LS mo 0 | T3: 10-1074 + VRC07-523LS | T4: PGT121 + PGDM1400 + VRC07-523LS mo(0, 4)
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/6 | 0/6 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/6 | 0/6 | 0/9
Other Adverse Events (participants affected / at risk) | 5/6 | 6/6 | 4/6 | 4/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T1: PGT121 + VRC07-523LS mo 0 (N=6) | T2: PGDM1400 + VRC07-523LS mo 0 (N=6) | T3: 10-1074 + VRC07-523LS (N=6) | T4: PGT121 + PGDM1400 + VRC07-523LS mo(0, 4) (N=9)
Any Event in SOC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T1: PGT121 + VRC07-523LS mo 0 (N=6) | T2: PGDM1400 + VRC07-523LS mo 0 (N=6) | T3: 10-1074 + VRC07-523LS (N=6) | T4: PGT121 + PGDM1400 + VRC07-523LS mo(0, 4) (N=9)
Any Event in SOC (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Any Event in SOC (General disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Infections and infestations) | 3 (3) | 2 (2) | 1 (1) | 3 (3)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Latent tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal chlamydia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Any Event in SOC (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Investigations) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Any Event in SOC (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Any Event in SOC (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Androgenetic alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/21/NCT03928821/Prot_SAP_001.pdf
  • Informed Consent Form (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/21/NCT03928821/ICF_000.pdf